CLINICAL TRIAL: NCT02991859
Title: An Escalating Dose, Randomized, Placebo-controlled, Incomplete-block, 2-period Cross-over Study to Assess the Dose Response for Topical Efficacy Via Airway Responsiveness to Adenosine-5'-Monophosphate (AMP) Challenge and the Dose Response for Systemic Activity Via 24h Plasma Cortisol Suppression and Thereby the Relative Therapeutic Index for Fluticasone Furoate (FF), Fluticasone Propionate (FP) and Budesonide (BUD) in Asthmatic Subjects
Brief Title: Phase 2a, AMP Challenge, Dose Escalation Study to Assess the Dose Response for Topical Efficacy and Systemic Activity in Asthmatic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 203162; 2016-003002-14 (EudraCT Number)
Record Dates: First submitted 2016-12-09; First posted 2016-12-14 (Estimated); Results first posted 2020-03-30 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Asthma
Keywords: Dose-response; AMP challenge; cortisol suppression; dose escalation; therapeutic index
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; Dry Powder Inhalers; Fluticasone; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Arm AB - FF followed by FP (Experimental): Each treatment period (TP) comprises of 5 consecutive 7-day dosing phases with escalating doses of either FF or FP. In TP 1, subjects will receive evening (PM) dose of 1 puff of FF 25 microgram (mcg) (Total daily dose [TDD] = 25 mcg) in first phase followed by PM dose of 1 puff of FF 100 mcg (TDD = 100 mcg) in second phase; PM dose of 1 puff of FF 200 mcg (TDD = 200 mcg) in third phase; PM dose of 2 puff of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puff of FF 200 mcg (TDD = 800 mcg) in fifth phase. In TP 2, subjects will receive PM dose of 1 puff of FP 50 mcg (TDD = 50 mcg) in first phase followed by morning (AM) and PM doses of 1 puff each of FP 100 mcg (TDD = 200 mcg) in second phase; AM and PM doses of 1 puff each of FP 250 mcg (TDD = 500 mcg) in third phase; AM and PM doses of 1 puff each of FP 500 mcg (TDD = 1000 mcg) in fourth phase and AM and PM doses of 2 puffs each of FP 500 mcg (TDD = 2000 mcg) in fifth phase. Washout period will be of 25-42 days.
  Interventions: Drug: Fluticasone furoate (FF) Dry Powder Inhaler; Drug: Fluticasone propionate (FP) Dry Powder Inhaler
- Arm AC - FF followed by BUD (Experimental): Each TP comprises of 5 consecutive 7-day dosing phases with escalating doses of either FF or BUD. In TP 1, subjects will receive PM dose of 1 puff of FF 25 mcg (TDD = 25 mcg) in first phase followed by PM dose of 1 puff of FF 100 mcg (TDD = 100 mcg) in second phase; PM dose of 1 puff of FF 200 mcg (TDD = 200 mcg) in third phase; PM dose of 2 puffs of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puffs of FF 200 mcg (TDD = 800 mcg) in fifth phase. In TP 2, subjects will receive PM dose of 1 puff of BUD 100 mcg (TDD = 100 mcg) in first phase followed by AM and PM doses of 1 puff each of BUD 200 mcg (TDD = 400 mcg) in second phase; AM and PM doses of 1 puff each of BUD 400 mcg (TDD = 800 mcg) in third phase; AM and PM doses of 2 puffs each of BUD 400 mcg (TDD = 1600 mcg) in fourth phase and AM and PM doses of 4 puffs each of BUD 400 mcg (TDD = 3200 mcg) in fifth phase. Washout period will be of 25-42 days.
  Interventions: Drug: Fluticasone furoate (FF) Dry Powder Inhaler; Drug: Budesonide (BUD) Turbuhaler
- Arm AD - FF followed by ELLIPTA Placebo (Experimental): Each TP comprises of 5 consecutive 7-day dosing phases with escalating doses of either FF or ELLIPTA Placebo. In TP 1, subjects will receive PM dose of 1 puff of FF 25 mcg (TDD = 25 mcg) in first phase followed by PM dose of 1 puff of FF 100 mcg (TDD = 100 mcg) in second phase; PM dose of 1 puff of FF 200 mcg (TDD = 200 mcg) in third phase; PM dose of 2 puffs of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puffs of FF 200 mcg (TDD = 800 mcg) in fifth phase. In TP 2, subjects will receive PM dose of 1 puff of ELLIPTA Placebo in first, second and third phases followed by PM dose of 2 puffs of ELLIPTA Placebo in fourth phase and PM dose of 4 puffs of ELLIPTA Placebo in fifth phase. Washout period will be of 25-42 days.
  Interventions: Drug: Fluticasone furoate (FF) Dry Powder Inhaler; Drug: Placebo (ELLIPTA or DISKUS)
- Arm BA - FP followed by FF (Experimental): Each TP comprises of 5 consecutive 7-day dosing phases with escalating doses of either FP or FF. In TP 1, subjects will receive PM dose of 1 puff of FP 50 mcg (TDD = 50 mcg) in first phase followed by AM and PM doses of 1 puff each of FP 100 mcg (TDD = 200 mcg) in second phase; AM and PM doses of 1 puff each of FP 250 mcg (TDD = 500 mcg) in third phase; AM and PM doses of 1 puff each of FP 500 mcg (TDD = 1000 mcg) in fourth phase and AM and PM doses of 2 puffs each of FP 500 mcg (TDD = 2000 mcg) in fifth phase. In TP 2, subjects will receive PM dose of 1 puff of FF 25 mcg (TDD = 25 mcg) in first phase followed by PM dose of 1 puff of FF 100 mcg (TDD = 100 mcg) in second phase; PM dose of 1 puff of FF 200 mcg (TDD = 200 mcg) in third phase; PM dose of 2 puffs of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puffs of FF 200 mcg (TDD = 800 mcg) in fifth phase. Washout period will be of 25-42 days.
  Interventions: Drug: Fluticasone furoate (FF) Dry Powder Inhaler; Drug: Fluticasone propionate (FP) Dry Powder Inhaler
- Arm BC - FP followed by BUD (Experimental): Each TP comprises of 5 consecutive 7-day dosing phases with escalating doses of either FP or BUD. In TP 1, subjects will receive PM dose of 1 puff of FP 50 mcg (TDD = 50 mcg) in first phase followed by AM and PM doses of 1 puff each of FP 100 mcg (TDD = 200 mcg) in second phase; AM and PM doses of 1 puff each of FP 250 mcg (TDD = 500 mcg) in third phase; AM and PM doses of 1 puff each of FP 500 mcg (TDD = 1000 mcg) in fourth phase and AM and PM doses of 2 puffs each of FP 500 mcg (TDD = 2000 mcg) in fifth phase. In TP 2, subjects will receive PM dose of 1 puff of BUD 100 mcg (TDD =100 mcg) in first phase followed by AM and PM doses of 1 puff each of BUD 200 mcg (TDD = 400 mcg) in second phase; AM and PM doses of 1 puff each of BUD 400 mcg (TDD = 800 mcg) in third phase; AM and PM doses of 2 puffs each of BUD 400 mcg (TDD =1600 mcg) in fourth phase and AM and PM doses of 4 puffs each of BUD 400 mcg (TDD = 3200 mcg) in fifth phase. Washout period will be of 25-42 days.
  Interventions: Drug: Fluticasone propionate (FP) Dry Powder Inhaler; Drug: Budesonide (BUD) Turbuhaler
- Arm BE - FP followed by DISKUS Placebo (Experimental): Each TP comprises of 5 consecutive 7-day dosing phases with escalating doses of either FP or DISKUS Placebo. In TP 1, subjects will receive PM dose of 1 puff of FP 50 mcg (TDD = 50 mcg) in first phase followed by AM and PM doses of 1 puff each of FP 100 mcg (TDD = 200 mcg) in second phase; AM and PM doses of 1 puff each of FP 250 mcg (TDD = 500 mcg) in third phase; AM and PM doses of 1 puff each of FP 500 mcg (TDD = 1000 mcg) in fourth phase and AM and PM doses of 2 puffs each of FP 500 mcg (TDD = 2000 mcg) in fifth phase. In TP 2, subjects will receive PM dose of 1 puff of DISKUS Placebo in first phase followed by AM and PM doses of 1 puff each DISKUS Placebo in second, third and fourth phase; AM and PM doses of 2 puffs each of DISKUS Placebo in fifth phase. Each TP will be followed by a washout period of 25-42 days.
  Interventions: Drug: Fluticasone propionate (FP) Dry Powder Inhaler; Drug: Placebo (ELLIPTA or DISKUS)
- Arm CA - BUD followed by FF (Experimental): Each TP comprises of 5 consecutive 7-day dosing phases with escalating doses of either BUD or FF. In TP 1, subjects will receive PM dose of 1 puff of BUD 100 mcg (TDD =100 mcg) in first phase followed by AM and PM doses of 1 puff each of BUD 200 mcg (TDD =400 mcg) in second phase; AM and PM doses of 1 puff each of BUD 400 mcg (TDD = 800 mcg) in third phase; AM and PM doses of 2 puffs each of BUD 400 mcg (TDD =1600 mcg) in fourth phase and AM and PM doses of 4 puffs each of BUD 400 mcg (TDD = 3200 mcg) in fifth phase. In TP 2, subjects will receive PM dose of 1 puff of FF 25 mcg (TDD = 25 mcg) in first phase followed by PM dose of 1 puff of FF 100 mcg (TDD = 100 mcg) in second phase; PM dose of 1 puff of FF 200 mcg (TDD = 200 mcg) in third phase; PM dose of 2 puffs of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puffs of FF 200 mcg (TDD = 800 mcg) in fifth phase. Washout period will be of 25-42 days.
  Interventions: Drug: Fluticasone furoate (FF) Dry Powder Inhaler; Drug: Budesonide (BUD) Turbuhaler
- Arm CB - BUD followed by FP (Experimental): Each TP comprises of 5 consecutive 7-day dosing phases with escalating doses of either BUD or FP. In TP 1, subjects will receive PM dose of 1 puff of BUD 100 mcg (TDD =100 mcg) in first phase followed by AM and PM doses of 1 puff each of BUD 200 mcg (TDD =400 mcg) in second phase; AM and PM doses of 1 puff each of BUD 400 mcg (TDD = 800 mcg) in third phase; AM and PM doses of 2 puffs each of BUD 400 mcg (TDD =1600 mcg) in fourth phase and AM and PM doses of 4 puffs each of BUD 400 mcg (TDD = 3200 mcg) in fifth phase. In TP 2, subjects will receive PM dose of 1 puff of FP 50 mcg (TDD = 50 mcg) in first phase followed by AM and PM doses of 1 puff each of FP 100 mcg (TDD = 200 mcg) in second phase; AM and PM doses of 1 puff each of FP 250 mcg (TDD =500 mcg) in third phase; AM and PM doses of 1 puff each of FP 500 mcg (TDD = 1000 mcg) in fourth phase and AM and PM doses of 2 puffs each of FP 500 mcg (TDD = 2000 mcg) in fifth phase. Washout period will be of 25-42 days.
  Interventions: Drug: Fluticasone propionate (FP) Dry Powder Inhaler; Drug: Budesonide (BUD) Turbuhaler
- Arm CE - BUD followed by DISKUS Placebo (Experimental): Each TP comprises of 5 consecutive 7-day dosing phases with escalating doses of either BUD or DISKUS Placebo. In TP 1, subjects will receive PM dose of 1 puff of BUD 100 mcg (TDD =100 mcg) in first phase followed by AM and PM doses of 1 puff each of BUD 200 mcg (TDD =400 mcg) in second phase; AM and PM doses of 1 puff each of BUD 400 mcg (TDD = 800 mcg) in third phase; AM and PM doses of 2 puffs each of BUD 400 mcg (TDD =1600 mcg) in fourth phase and AM and PM doses of 4 puffs each of BUD 400 mcg (TDD = 3200 mcg) in fifth phase. In TP 2, subjects will receive PM dose of 1 puff of DISKUS Placebo in first phase followed by AM and PM doses of 1 puff each DISKUS Placebo in second, third and fourth phase; and AM and PM doses of 2 puffs each of DISKUS Placebo in fifth phase. Washout period will be of 25-42 days.
  Interventions: Drug: Budesonide (BUD) Turbuhaler; Drug: Placebo (ELLIPTA or DISKUS)
- Arm DA - ELLIPTA Placebo followed by FF (Experimental): Each TP comprises of 5 consecutive 7-day dosing phases with escalating doses of either ELLIPTA Placebo or FF. In TP 1, subjects will receive PM dose of 1 puff of ELLIPTA Placebo in first, second and third phase followed by PM dose of 2 puffs of ELLIPTA Placebo in fourth phase and PM dose of 4 puffs of ELLIPTA Placebo in fifth phase. In TP 2, subjects will receive PM dose of 1 puff of FF 25 mcg (TDD = 25 mcg) in first phase followed by PM dose of 1 puff of FF 100 mcg (TDD = 100 mcg) in second phase; PM dose of 1 puff of FF 200 mcg (TDD = 200 mcg) in third phase; PM dose of 2 puffs of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puffs of FF 200 mcg (TDD = 800 mcg) in fifth phase. Washout period will be of 25-42 days.
  Interventions: Drug: Fluticasone furoate (FF) Dry Powder Inhaler; Drug: Placebo (ELLIPTA or DISKUS)
- Arm EB - DISKUS Placebo followed by FP (Experimental): Each TP comprises of 5 consecutive 7-day dosing phases with escalating doses of either DISKUS Placebo or FP. TP 1, subjects will receive PM dose of 1 puff of DISKUS Placebo in first phase followed by AM and PM doses of 1 puff each of DISKUS Placebo in second, third and fourth phase; AM and PM doses of 2 puffs each of DISKUS Placebo in fifth phase. In TP 2, subjects will receive PM dose of 1 puff of FP 50 mcg (TDD = 50 mcg) in first phase followed by AM and PM doses of 1 puff each of FP 100 mcg (TDD = 200 mcg) in second phase; AM and PM doses of 1 puff each of FP 250 mcg (TDD = 500 mcg) in third phase; AM and PM doses of 1 puff each of FP 500 mcg (TDD = 1000 mcg) in fourth phase and AM and PM doses of 2 puffs each of FP 500 mcg (TDD = 2000 mcg) in fifth phase. Washout period will be of 25-42 days.
  Interventions: Drug: Fluticasone propionate (FP) Dry Powder Inhaler; Drug: Placebo (ELLIPTA or DISKUS)
- Arm DC - ELLIPTA Placebo followed by BUD (Experimental): Each TP comprises of 5 consecutive 7-day dosing phases with escalating doses of either ELLIPTA Placebo or BUD. In TP 1, subjects will receive PM dose of 1 puff of ELLIPTA Placebo in first, second and third phase followed by PM dose of 2 puffs of ELLIPTA Placebo in fourth phase and PM dose of 4 puffs of ELLIPTA Placebo in fifth phase. In TP 2, subjects will receive PM dose of 1 puff of BUD 100 mcg (TDD =100 mcg) in first phase followed by AM and PM doses of 1 puff each of BUD 200 mcg (TDD =400 mcg) in second phase; AM and PM doses of 1 puff each of BUD 400 mcg (TDD = 800 mcg) in third phase; AM and PM doses of 2 puffs each of BUD 400 mcg (TDD =1600 mcg) in fourth phase and AM and PM doses of 4 puffs each of BUD 400 mcg (TDD = 3200 mcg) in fifth phase. Washout period will be of 25-42 days.
  Interventions: Drug: Budesonide (BUD) Turbuhaler; Drug: Placebo (ELLIPTA or DISKUS)

INTERVENTIONS:
Drug: Fluticasone furoate (FF) Dry Powder Inhaler — Dry inhalation powder 25 mcg, 100 mcg, and 200 mcg per blister strip will be administered using ELLIPTA for both treatment periods
  Arms: Arm AB - FF followed by FP; Arm AC - FF followed by BUD; Arm AD - FF followed by ELLIPTA Placebo; Arm BA - FP followed by FF; Arm CA - BUD followed by FF; Arm DA - ELLIPTA Placebo followed by FF
Drug: Fluticasone propionate (FP) Dry Powder Inhaler — Dry Inhalation powder 50 mcg, 100 mcg, 250 mcg, and 500 mcg per blister strip will be administered using DISKUS for both treatment periods
  Arms: Arm AB - FF followed by FP; Arm BA - FP followed by FF; Arm BC - FP followed by BUD; Arm BE - FP followed by DISKUS Placebo; Arm CB - BUD followed by FP; Arm EB - DISKUS Placebo followed by FP
Drug: Budesonide (BUD) Turbuhaler — Budesonide comprises white to off-white rounded granules, which disintegrate to a fine powder upon slight pressure, will be administered using Turbuhaler for both treatment periods.
  Arms: Arm AC - FF followed by BUD; Arm BC - FP followed by BUD; Arm CA - BUD followed by FF; Arm CB - BUD followed by FP; Arm CE - BUD followed by DISKUS Placebo; Arm DC - ELLIPTA Placebo followed by BUD
Drug: Placebo (ELLIPTA or DISKUS) — Lactose dry powder inhaler will be administered using ELLIPTA or DISKUS for both treatment periods.
  Arms: Arm AD - FF followed by ELLIPTA Placebo; Arm BE - FP followed by DISKUS Placebo; Arm CE - BUD followed by DISKUS Placebo; Arm DA - ELLIPTA Placebo followed by FF; Arm DC - ELLIPTA Placebo followed by BUD; Arm EB - DISKUS Placebo followed by FP

SUMMARY:
This is a randomized, placebo-controlled, 2-period crossover, escalating repeat dose study, aiming to investigate whether higher potency of different inhaled corticosteroid confers an improvement in the topical efficacy to systemic activity ratio in asthmatic subjects. It will compare the dose response for topical efficacy via airway responsiveness (to adenosine-5'-monophosphate [AMP] challenge), and the dose response for systemic activity via 24 hour plasma cortisol suppression, and thereby compare the relative therapeutic index, for the following inhaled corticosteroids: fluticasone furoate (FF), fluticasone propionate (FP) and budesonide (BUD). There will be a screening visit 4 - 42 days before the first dose of study treatment, and AMP challenge Provocative concentration 20 (PC20) of <=80 milligrams per milliliter (mg/mL) at screening visit 2 i.e. at 4 - 14 days before the first dose of study treatment. Subjects will be randomized to one of 5 or 12 treatment sequences, and will have one or two treatment periods, each comprising 5 consecutive 7-day phases of escalating doses of either FF, FP, BUD or placebo. There will be a 25- to 42-day washout period between treatment periods. The study duration for each subject will be approximately 13 or 24 weeks including the follow-up period.

ELIGIBILITY:
Inclusion Criteria - Subjects must be 18 to 65 years of age inclusive, at the time of signing the informed Consent. - Documented history of bronchial asthma, first diagnosed at least 6 months prior to the screening visit - Pre-bronchodilator FEV1 >=65% of predicted at screening; the pre-dose baseline FEV1 should not have changed significantly in the opinion of the investigator from the screening baseline value and should be >=65% predicted for the subject to continue - Documented sensitivity to AMP with a provocative concentration of AMP resulting in a fall of >=20% FEV1 with a PC20 AMP <=80 mg/mL at the screening visit - Current therapy could include short-acting Beta2-agonists (SABA) prescribed SABA for at least 12 weeks prior to screening, if needed; subjects receiving low-dose ICS may take part after a 4-week ICS washout prior to AMP challenge. The subject's asthma symptoms must remain stable during this 4-week period as assessed at screening visit 2. Stable asthma is defined as no more than 2 consecutive days where >=12 inhalations/day of salbutamol were used; or no severe asthma exacerbations requiring use of systemic corticosteroids (tablets, suspension, or injection) or an in-patient hospitalization or emergency department visit due to asthma that required systemic corticosteroids; or no clinical asthma worsening which in the opinion of the investigator requires additional asthma treatment other than study medication or salbutamol; subjects taking Long-acting beta2-agonist (LABA), long-acting muscarinic antagonist (LAMA), leukotriene receptor antagonist (LTRA) therapy within three months prior to the start of the study are not eligible; subjects taking biological therapies within 6 months prior to start of the study are not eligible. - Bodyweight >=50 Kilogram (kg) and BMI within the range 18.0-35.0 kg/meter (m)^2 (inclusive) - Male and female. Females: A female subject is eligible to participate if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [HCG] test), not lactating, and at least one of the following conditions applies prior to randomization: • Non-reproductive potential defined as pre-menopausal females with one of the following: Documented tubal ligation; Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion; Hysterectomy; Documented Bilateral Oophorectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea, in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment. • Reproductive potential and agrees to follow one of the highly effective methods for avoiding pregnancy in females of reproductive potential from 30 days prior to the first dose of study medication and until at least five terminal half-lives after the last dose of study medication. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception. - Aspartate aminotransferase and Alanine transaminase <2x upper limit of normal (ULN); alkaline phosphatase and bilirubin ≤1.5 x ULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%) - Light smokers, who smoke <=20 cigarettes per week or equivalent unit dose of other tobacco products or e-cigarettes, are eligible for the study. Smokers who intend to stop, reduce or increase their smoking habit during the study period are not eligible. - Having provided written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria: - A history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures within the last 5 years. - Other significant pulmonary diseases to include (but not limited to) severe pneumonia within 6 months of the screening visit, pneumothorax, atelectasis, pulmonary fibrotic disease, bronchopulmonary dysplasia, chronic bronchitis, emphysema, chronic obstructive pulmonary disease, tuberculosis or other respiratory abnormalities other than asthma. - Culture-documented or suspected bacterial or viral infection of the upper or lower respiratory tract, sinus or middle ear within 4 weeks of screening that: In the opinion of the investigator, is expected to affect the subject's asthma status or the subject's ability to participate in the study. - A subject will not be eligible if he/she has clinical visual evidence of oral candidiasis at screening. - Any asthma exacerbation requiring oral corticosteroids within 12 weeks of screening or that resulted in overnight hospitalization requiring additional treatment for asthma within 6 months prior to randomization. - Use of prohibited medications including, anti-depressant drugs, and anti-asthma drugs (other than short acting inhaled beta-agonists supplied as rescue medication, oral contraceptives, non-steroidal anti-inflammatory drugs, stable doses of antihistamines, and paracetamol) for 1 week prior to screening and throughout the course of the study. Anti-histamines should be withheld 4 days prior to AMP challenge; subjects must also be able to abstain from short acting inhaled beta-agonists, for 8 hours prior to spirometry. - Subjects undergoing de-sensitization therapy - Current smokers who smoke > 20 cigarettes per week or the equivalent unit dose of other tobacco products or e-cigarettes, or smokers with a smoking history of >=10 pack years. - History of regular alcohol consumption exceeding 21 units per week for men and 14 units per week for females (1 unit =5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of spirits) within 6 months of screening. - All subjects who are currently or in the last month have worked night-shifts are excluded from the study - Exposure to more than four new chemical entities within 12 months prior to the first dosing day or received an investigational product within 30 days of study start, or 5 half-lives of study drug if that is longer. - A subject has any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the study results if the condition/disease exacerbated during the study. (e.g. stroke or myocardial infarction within 3 months, uncontrolled hypertension, congestive heart failure, uncontrolled diabetes mellitus.) - Evidence of cancer or history of cancer in the past 5 years other than adequately treated basal or squamous cell carcinoma of the skin or adequately treated in situ carcinoma of the cervix. - Pregnant females as determined by positive urine HCG test at screening or by positive urine HCG test prior to dosing and lactating females. - Subjects with active or chronic infections including hepatitis B or C, human immunodeficiency virus. A positive serology at screening. - Allergies: History of severe milk protein allergy Drug Allergy defined as any adverse reaction including immediate or delayed hypersensitivity to intranasal, inhaled, or systemic corticosteroid therapy. Known or suspected sensitivity to the constituents of FF, FP or BUD (i.e., lactose or magnesium stearate etc.) Historical Allergy defined as history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation. - Significant abnormality in the 12-lead electrocardiogram (ECG) performed at screening. The mean of the three individual ECGs will be taken. Mean QT interval corrected for heart rate (QTc) >450 millisecond (msec) for males or QTc>470 msec for female subjects and >480 in subjects with bundle branch block. The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- GSK Investigational Site, Berlin, Germany
- United Kingdom (2):
  - GSK Investigational Site, Harrow, Middlesex
  - GSK Investigational Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20386

REFERENCES:
- [Derived] Daley-Yates P, Brealey N, Thomas S, Austin D, Shabbir S, Harrison T, Singh D, Barnes N. Therapeutic index of inhaled corticosteroids in asthma: A dose-response comparison on airway hyperresponsiveness and adrenal axis suppression. Br J Clin Pharmacol. 2021 Feb;87(2):483-493. doi: 10.1111/bcp.14406. Epub 2020 Jun 17. PMID 32484940

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 56 participants were enrolled across 1 center in Germany and 2 centers in the United Kingdom.
Pre-assignment Details: A total of 165 participants were screened of which 109 failed screening and 56 participants were enrolled in study. Of the 56 participants enrolled,only 54 were randomized and received at least one dose of study medication. Only 7 participants were withdrawn from the study, 2 participants who were not withdrawn, entered Period 2 esc Phase 1.
Groups:
- Arm AB - FF Followed by FP: Participants received evening (PM) dose of 1 puff of Fluticasone Furoate (FF) 25 microgram (mcg) (Total daily dose [TDD] = 25 mcg) in first dose escalation phase followed by PM dose of 1 puff of FF 100 mcg (TDD = 100 mcg) in second phase; PM dose of 1 puff of FF 200 mcg (TDD = 200 mcg) in third phase; PM dose of 2 puff of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puff of FF 200 mcg (TDD = 800 mcg) in fifth phase. In TP 2, participants received PM dose of 1 puff of FP 50 mcg (TDD = 50 mcg) in first phase followed by morning (AM) and PM doses of 1 puff each of FP 100 mcg (TDD = 200 mcg) in second phase; AM and PM doses of 1 puff each of FP 250 mcg (TDD = 500 mcg) in third phase; AM and PM doses of 1 puff each of FP 500 mcg (TDD = 1000 mcg) in fourth phase and AM and PM doses of 2 puffs each of FP 500 mcg (TDD = 2000 mcg) in fifth phase. Washout period was of 25-42 days.
- Arm AC - FF Followed by BUD: Participants received PM dose of 1 puff of FF 25mcg (TDD=25 mcg) in first phase followed by PM dose of 1 puff of FF 100 mcg (TDD=100 mcg) in second phase; PM dose of 1 puff of FF 200mcg (TDD=200 mcg) in third phase; PM dose of 2 puffs of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puffs of FF 200 mcg (TDD =800 mcg) in fifth phase. In TP 2, participants received PM dose of 1 puff of BUD 100 mcg (TDD=100 mcg) in first phase followed by AM and PM doses of 1 puff each of BUD 200 mcg (TDD=400 mcg) in second phase; AM and PM doses of 1 puff each of BUD 400 mcg (TDD=800 mcg) in third phase; AM and PM doses of 2 puffs each of BUD 400 mcg (TDD=1600 mcg) in fourth phase and AM and PM doses of 4 puffs each of BUD 400 mcg (TDD=3200 mcg) in fifth phase. Washout period was of 25-42 days.
- Arm AD - FF Followed by ELLIPTA Placebo: Participants received PM dose of 1 puff of FF 25 mcg (TDD = 25 mcg) in first phase followed by PM dose of 1 puff of FF 100 mcg (TDD = 100 mcg) in second phase; PM dose of 1 puff of FF 200 mcg (TDD = 200 mcg) in third phase; PM dose of 2 puffs of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puffs of FF 200 mcg (TDD = 800 mcg) in fifth phase. In TP 2, participants received PM dose of 1 puff of ELLIPTA Placebo in first, second and third phases followed by PM dose of 2 puffs of ELLIPTA Placebo in fourth phase and PM dose of 4 puffs of ELLIPTA Placebo in fifth phase. Washout period was of 25-42 days.
- Arm BA - FP Followed by FF: Participants received PM dose of 1 puff of FP 50 mcg (TDD = 50 mcg) in first phase followed by AM and PM doses of 1 puff each of FP 100 mcg (TDD = 200 mcg) in second phase; AM and PM doses of 1 puff each of FP 250 mcg (TDD = 500 mcg) in third phase; AM and PM doses of 1 puff each of FP 500 mcg (TDD = 1000 mcg) in fourth phase and AM and PM doses of 2 puffs each of FP 500 mcg (TDD = 2000 mcg) in fifth phase. In TP 2, participants received PM dose of 1 puff of FF 25 mcg (TDD = 25 mcg) in first phase followed by PM dose of 1 puff of FF 100 mcg (TDD = 100 mcg) in second phase; PM dose of 1 puff of FF 200 mcg (TDD = 200 mcg) in third phase; PM dose of 2 puffs of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puffs of FF 200 mcg (TDD = 800 mcg) in fifth phase. Washout period was of 25-42 days.
- Arm BC - FP Followed by BUD: Participants received PM dose of 1 puff of FP 50 mcg (TDD = 50 mcg) in first phase followed by AM and PM doses of 1 puff each of FP 100 mcg (TDD = 200 mcg) in second phase; AM and PM doses of 1 puff each of FP 250 mcg (TDD = 500 mcg) in third phase; AM and PM doses of 1 puff each of FP 500 mcg (TDD = 1000 mcg) in fourth phase and AM and PM doses of 2 puffs each of FP 500 mcg (TDD = 2000 mcg) in fifth phase. In TP 2, participants received PM dose of 1 puff of BUD 100 mcg (TDD =100 mcg) in first phase followed by AM and PM doses of 1 puff each of BUD 200 mcg (TDD = 400 mcg) in second phase; AM and PM doses of 1 puff each of BUD 400 mcg (TDD = 800 mcg) in third phase; AM and PM doses of 2 puffs each of BUD 400 mcg (TDD =1600 mcg) in fourth phase and AM and PM doses of 4 puffs each of BUD 400 mcg (TDD = 3200 mcg) in fifth phase. Washout period was of 25-42 days.
- Arm BE - FP Followed by DISKUS Placebo: Participants received PM dose of 1 puff of FP 50 mcg (TDD = 50 mcg) in first phase followed by AM and PM doses of 1 puff each of FP 100 mcg (TDD = 200 mcg) in second phase; AM and PM doses of 1 puff each of FP 250 mcg (TDD = 500 mcg) in third phase; AM and PM doses of 1 puff each of FP 500 mcg (TDD = 1000 mcg) in fourth phase and AM and PM doses of 2 puffs each of FP 500 mcg (TDD = 2000 mcg) in fifth phase. In TP 2, participants received PM dose of 1 puff of DISKUS Placebo in first phase followed by AM and PM doses of 1 puff each DISKUS Placebo in second, third and fourth phase; AM and PM doses of 2 puffs each of DISKUS Placebo in fifth phase. Washout period was of 25-42 days.
- Arm CA - BUD Followed by FF: Participants received PM dose of 1 puff of BUD 100 mcg (TDD =100 mcg) in first phase followed by AM and PM doses of 1 puff each of BUD 200 mcg (TDD =400 mcg) in second phase; AM and PM doses of 1 puff each of BUD 400 mcg (TDD = 800 mcg) in third phase; AM and PM doses of 2 puffs each of BUD 400 mcg (TDD =1600 mcg) in fourth phase and AM and PM doses of 4 puffs each of BUD 400 mcg (TDD = 3200 mcg) in fifth phase. In TP 2, participants received PM dose of 1 puff of FF 25 mcg (TDD = 25 mcg) in first phase followed by PM dose of 1 puff of FF 100 mcg (TDD = 100 mcg) in second phase; PM dose of 1 puff of FF 200 mcg (TDD = 200 mcg) in third phase; PM dose of 2 puffs of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puffs of FF 200 mcg (TDD = 800 mcg) in fifth phase. Washout period was of 25-42 days.
- Arm CB - BUD Followed by FP: Participants received PM dose of 1 puff of BUD 100 mcg (TDD =100 mcg) in first phase followed by AM and PM doses of 1 puff each of BUD 200 mcg (TDD =400 mcg) in second phase; AM and PM doses of 1 puff each of BUD 400 mcg (TDD = 800 mcg) in third phase; AM and PM doses of 2 puffs each of BUD 400 mcg (TDD =1600 mcg) in fourth phase and AM and PM doses of 4 puffs each of BUD 400 mcg (TDD = 3200 mcg) in fifth phase. In TP 2, participants received PM dose of 1 puff of FP 50 mcg (TDD = 50 mcg) in first phase followed by AM and PM doses of 1 puff each of FP 100 mcg (TDD = 200 mcg) in second phase; AM and PM doses of 1 puff each of FP 250 mcg (TDD =500 mcg) in third phase; AM and PM doses of 1 puff each of FP 500 mcg (TDD = 1000 mcg) in fourth phase and AM and PM doses of 2 puffs each of FP 500 mcg (TDD = 2000 mcg) in fifth phase. Washout period was of 25-42 days.
- Arm CE - BUD Followed by DISKUS Placebo: Participants received PM dose of 1 puff of BUD as 100 mcg in first phase followed by BUD 200 mcg 1 puff AM and PM (TDD=400 mcg), in third phase BUD 400 mcg 1 puff AM and PM (TDD=800 mcg) followed by BUD 400 mcg 2 puffs AM and PM(TDD=1600mcg) in fourth phase followed by BUD 400 mcg 4puffs AM and PM (TDD=3200mcg) in TP1. In TP 2 participants received DISKUS placebo 1 puff PM in first phase followed by DISKUS placebo 1 puff AM and PM in second phase followed by DISKUS placebo 1 puff AM and PM in third phase followed by DISKUS placebo 1 puff AM and PM in fourth phase followed by DISKUS placebo 2 puffs AM and PM in fifth phase. Washout period was of 25-42 days.
- Arm DA - ELLIPTA Placebo Followed by FF: Participants received PM dose of 1 puff of ELLIPTA Placebo in first, second and third phase followed by PM dose of 2 puffs of ELLIPTA Placebo in fourth phase and PM dose of 4 puffs of ELLIPTA Placebo in fifth phase. In TP 2, participants will receive PM dose of 1 puff of FF 25 mcg (TDD = 25 mcg) in first phase followed by PM dose of 1 puff of FF 100 mcg (TDD = 100 mcg) in second phase; PM dose of 1 puff of FF 200 mcg (TDD = 200 mcg) in third phase; PM dose of 2 puffs of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puffs of FF 200 mcg (TDD = 800 mcg) in fifth phase. Washout period was of 25-42 days.
- EB - DISKUS Placebo Followed by FP: Participants received PM dose of 1 puff of DISKUS Placebo in first phase followed by AM and PM doses of 1 puff each of DISKUS Placebo in second, third and fourth phase; AM and PM doses of 2 puffs each of DISKUS Placebo in fifth phase. In TP 2, participants received PM dose of 1 puff of FP 50 mcg (TDD = 50 mcg) in first phase followed by AM and PM doses of 1 puff each of FP 100 mcg (TDD = 200 mcg) in second phase; AM and PM doses of 1 puff each of FP 250 mcg (TDD = 500 mcg) in third phase; AM and PM doses of 1 puff each of FP 500 mcg (TDD = 1000 mcg) in fourth phase and AM and PM doses of 2 puffs each of FP 500 mcg (TDD = 2000 mcg) in fifth phase. Washout period was of 25-42 days.
- Arm DC - ELLIPTA Placebo Followed by BUD: Participants received PM dose of 1 puff of ELLIPTA Placebo in first, second and third phase followed by PM dose of 2 puffs of ELLIPTA Placebo in fourth phase and PM dose of 4 puffs of ELLIPTA Placebo in fifth phase. In TP 2, participants received PM dose of 1 puff of BUD 100 mcg (TDD =100 mcg) in first phase followed by AM and PM doses of 1 puff each of BUD 200 mcg (TDD =400 mcg) in second phase; AM and PM doses of 1 puff each of BUD 400 mcg (TDD = 800 mcg) in third phase; AM and PM doses of 2 puffs each of BUD 400 mcg (TDD =1600 mcg) in fourth phase and AM and PM doses of 4 puffs each of BUD 400 mcg (TDD = 3200 mcg) in fifth phase. Washout period was of 25-42 days.
- Fluticasone Furoate (FF): Participants received evening (PM) dose of 1 puff of FF 25 microgram (mcg) (Total daily dose [TDD] = 25 mcg) in first dose escalation phase followed by PM dose of 1 puff of FF 100 mcg (TDD = 100 mcg) in second phase; PM dose of 1 puff of FF 200 mcg (TDD = 200 mcg) in third phase; PM dose of 2 puff of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puff of FF 200 mcg (TDD = 800 mcg) in fifth phase.
- Fluticasone Propionate (FP): Participants received PM dose of 1 puff of FP 50 mcg (TDD = 50 mcg) in first phase followed by morning (AM) and PM doses of 1 puff each of FP 100 mcg (TDD = 200 mcg) in second phase; AM and PM doses of 1 puff each of FP 250 mcg (TDD = 500 mcg) in third phase; AM and PM doses of 1 puff each of FP 500 mcg (TDD = 1000 mcg) in fourth phase and AM and PM doses of 2 puffs each of FP 500 mcg (TDD = 2000 mcg) in fifth phase.
- Budesonide (BUD): Participants received PM dose of 1 puff of BUD 100 mcg (TDD=100 mcg) in first phase followed by AM and PM doses of 1 puff each of BUD 200 mcg (TDD=400 mcg) in second phase; AM and PM doses of 1 puff each of BUD 400 mcg (TDD=800 mcg) in third phase; AM and PM doses of 2 puffs each of BUD 400 mcg (TDD=1600 mcg) in fourth phase and AM and PM doses of 4 puffs each of BUD 400 mcg (TDD=3200 mcg) in fifth phase.
- ELLIPTA: Participants received PM dose of 1 puff of ELLIPTA Placebo in first, second and third phases followed by PM dose of 2 puffs of ELLIPTA Placebo in fourth phase and PM dose of 4 puffs of ELLIPTA Placebo in fifth phase.
- DISKUS: Participants received PM dose of 1 puff of DISKUS Placebo in first phase followed by AM and PM doses of 1 puff each DISKUS Placebo in second, third and fourth phase; AM and PM doses of 2 puffs each of DISKUS Placebo in fifth phase.
Period: Period 1,Escalation Phase 1,Upto Day 7
Arm/Group | Arm AB - FF Followed by FP | Arm AC - FF Followed by BUD | Arm AD - FF Followed by ELLIPTA Placebo | Arm BA - FP Followed by FF | Arm BC - FP Followed by BUD | Arm BE - FP Followed by DISKUS Placebo | Arm CA - BUD Followed by FF | Arm CB - BUD Followed by FP | Arm CE - BUD Followed by DISKUS Placebo | Arm DA - ELLIPTA Placebo Followed by FF | EB - DISKUS Placebo Followed by FP | Arm DC - ELLIPTA Placebo Followed by BUD | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD) | ELLIPTA | DISKUS
Started | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 | 6 | 3 | 3
Completed | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 | 6 | 3 | 3
Not Completed | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 1,Escalation Phase2,Upto Day 14
Arm/Group | Arm AB - FF Followed by FP | Arm AC - FF Followed by BUD | Arm AD - FF Followed by ELLIPTA Placebo | Arm BA - FP Followed by FF | Arm BC - FP Followed by BUD | Arm BE - FP Followed by DISKUS Placebo | Arm CA - BUD Followed by FF | Arm CB - BUD Followed by FP | Arm CE - BUD Followed by DISKUS Placebo | Arm DA - ELLIPTA Placebo Followed by FF | EB - DISKUS Placebo Followed by FP | Arm DC - ELLIPTA Placebo Followed by BUD | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD) | ELLIPTA | DISKUS
Started | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 | 6 | 3 | 3
Completed | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 | 6 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period1, Escalation Phase3, Upto Day21
Arm/Group | Arm AB - FF Followed by FP | Arm AC - FF Followed by BUD | Arm AD - FF Followed by ELLIPTA Placebo | Arm BA - FP Followed by FF | Arm BC - FP Followed by BUD | Arm BE - FP Followed by DISKUS Placebo | Arm CA - BUD Followed by FF | Arm CB - BUD Followed by FP | Arm CE - BUD Followed by DISKUS Placebo | Arm DA - ELLIPTA Placebo Followed by FF | EB - DISKUS Placebo Followed by FP | Arm DC - ELLIPTA Placebo Followed by BUD | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD) | ELLIPTA | DISKUS
Started | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 7 | 7 | 6 | 3 | 3
Completed | 2 | 2 | 2 | 2 | 2 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 6 | 6 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Period: Period1, Escalation Phase4, Upto Day28
Arm/Group | Arm AB - FF Followed by FP | Arm AC - FF Followed by BUD | Arm AD - FF Followed by ELLIPTA Placebo | Arm BA - FP Followed by FF | Arm BC - FP Followed by BUD | Arm BE - FP Followed by DISKUS Placebo | Arm CA - BUD Followed by FF | Arm CB - BUD Followed by FP | Arm CE - BUD Followed by DISKUS Placebo | Arm DA - ELLIPTA Placebo Followed by FF | EB - DISKUS Placebo Followed by FP | Arm DC - ELLIPTA Placebo Followed by BUD | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD) | ELLIPTA | DISKUS
Started | 2 | 2 | 2 | 2 | 2 | 2 (1 Par completed Phase 3 did not enter Phase 4) | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 6 | 6 | 3 | 3
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 6 | 6 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period1, Escalation Phase5, Upto Day35
Arm/Group | Arm AB - FF Followed by FP | Arm AC - FF Followed by BUD | Arm AD - FF Followed by ELLIPTA Placebo | Arm BA - FP Followed by FF | Arm BC - FP Followed by BUD | Arm BE - FP Followed by DISKUS Placebo | Arm CA - BUD Followed by FF | Arm CB - BUD Followed by FP | Arm CE - BUD Followed by DISKUS Placebo | Arm DA - ELLIPTA Placebo Followed by FF | EB - DISKUS Placebo Followed by FP | Arm DC - ELLIPTA Placebo Followed by BUD | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD) | ELLIPTA | DISKUS
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 (1 participant did not enter Esc Phase 5, and was not withdrawn) | 2 | 6 | 6 | 6 | 3 | 3
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 6 | 6 | 6 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash Out, Up to Day 77
Arm/Group | Arm AB - FF Followed by FP | Arm AC - FF Followed by BUD | Arm AD - FF Followed by ELLIPTA Placebo | Arm BA - FP Followed by FF | Arm BC - FP Followed by BUD | Arm BE - FP Followed by DISKUS Placebo | Arm CA - BUD Followed by FF | Arm CB - BUD Followed by FP | Arm CE - BUD Followed by DISKUS Placebo | Arm DA - ELLIPTA Placebo Followed by FF | EB - DISKUS Placebo Followed by FP | Arm DC - ELLIPTA Placebo Followed by BUD | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD) | ELLIPTA | DISKUS
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 0 (Participants did not enter washout and Period 2) | 0 (Participants did not enter washout and Period 2) | 0 (Participants did not enter washout and Period 2) | 0 (Participants did not enter washout and Period 2) | 0 (Participants did not enter washout and Period 2)
Completed | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period2, Escalation Phase1, Upto Day 84
Arm/Group | Arm AB - FF Followed by FP | Arm AC - FF Followed by BUD | Arm AD - FF Followed by ELLIPTA Placebo | Arm BA - FP Followed by FF | Arm BC - FP Followed by BUD | Arm BE - FP Followed by DISKUS Placebo | Arm CA - BUD Followed by FF | Arm CB - BUD Followed by FP | Arm CE - BUD Followed by DISKUS Placebo | Arm DA - ELLIPTA Placebo Followed by FF | EB - DISKUS Placebo Followed by FP | Arm DC - ELLIPTA Placebo Followed by BUD | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD) | ELLIPTA | DISKUS
Started | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 (1 Par directly entered into Period 2, Esc 1) | 2 (1 Par cont in P2 Esc 1 insteadP1 Esc 5, was not withdrawn) | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period2, Escalation Phase2, Upto Day 91
Arm/Group | Arm AB - FF Followed by FP | Arm AC - FF Followed by BUD | Arm AD - FF Followed by ELLIPTA Placebo | Arm BA - FP Followed by FF | Arm BC - FP Followed by BUD | Arm BE - FP Followed by DISKUS Placebo | Arm CA - BUD Followed by FF | Arm CB - BUD Followed by FP | Arm CE - BUD Followed by DISKUS Placebo | Arm DA - ELLIPTA Placebo Followed by FF | EB - DISKUS Placebo Followed by FP | Arm DC - ELLIPTA Placebo Followed by BUD | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD) | ELLIPTA | DISKUS
Started | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period2, Escalation Phase3, Upto Day 98
Arm/Group | Arm AB - FF Followed by FP | Arm AC - FF Followed by BUD | Arm AD - FF Followed by ELLIPTA Placebo | Arm BA - FP Followed by FF | Arm BC - FP Followed by BUD | Arm BE - FP Followed by DISKUS Placebo | Arm CA - BUD Followed by FF | Arm CB - BUD Followed by FP | Arm CE - BUD Followed by DISKUS Placebo | Arm DA - ELLIPTA Placebo Followed by FF | EB - DISKUS Placebo Followed by FP | Arm DC - ELLIPTA Placebo Followed by BUD | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD) | ELLIPTA | DISKUS
Started | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period2, Escalation Phase4, Upto Day 105
Arm/Group | Arm AB - FF Followed by FP | Arm AC - FF Followed by BUD | Arm AD - FF Followed by ELLIPTA Placebo | Arm BA - FP Followed by FF | Arm BC - FP Followed by BUD | Arm BE - FP Followed by DISKUS Placebo | Arm CA - BUD Followed by FF | Arm CB - BUD Followed by FP | Arm CE - BUD Followed by DISKUS Placebo | Arm DA - ELLIPTA Placebo Followed by FF | EB - DISKUS Placebo Followed by FP | Arm DC - ELLIPTA Placebo Followed by BUD | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD) | ELLIPTA | DISKUS
Started | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period2,Escalation Phase5,Upto Day 112
Arm/Group | Arm AB - FF Followed by FP | Arm AC - FF Followed by BUD | Arm AD - FF Followed by ELLIPTA Placebo | Arm BA - FP Followed by FF | Arm BC - FP Followed by BUD | Arm BE - FP Followed by DISKUS Placebo | Arm CA - BUD Followed by FF | Arm CB - BUD Followed by FP | Arm CE - BUD Followed by DISKUS Placebo | Arm DA - ELLIPTA Placebo Followed by FF | EB - DISKUS Placebo Followed by FP | Arm DC - ELLIPTA Placebo Followed by BUD | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD) | ELLIPTA | DISKUS
Started | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 1 | 2 | 2 | 1 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AC - FF Followed by BUD: Participants will receive PM dose of 1 puff of FF 25mcg (TDD=25 mcg) in first phase followed by PM dose of 1 puff of FF 100 mcg (TDD=100 mcg) in second phase; PM dose of 1 puff of FF 200mcg (TDD=200 mcg) in third phase; PM dose of 2 puffs of FF 200 mcg (TDD = 400 mcg) in fourth phase and PM dose of 4 puffs of FF 200 mcg (TDD =800 mcg) in fifth phase. In TP 2, participants will receive PM dose of 1 puff of BUD 100 mcg (TDD=100 mcg) in first phase followed by AM and PM doses of 1 puff each of BUD 200 mcg (TDD=400 mcg) in second phase; AM and PM doses of 1 puff each of BUD 400 mcg (TDD=800 mcg) in third phase; AM and PM doses of 2 puffs each of BUD 400 mcg (TDD=1600 mcg) in fourth phase and AM and PM doses of 4 puffs each of BUD 400 mcg (TDD=3200 mcg) in fifth phase. Washout period will be of 25-42 days
- Total: Total of all reporting groups
Arm/Group | Arm AB - FF Followed by FP | AC - FF Followed by BUD | Arm AD - FF Followed by ELLIPTA Placebo | Arm BA - FP Followed by FF | Arm BC - FP Followed by BUD | Arm BE - FP Followed by DISKUS Placebo | Arm CA - BUD Followed by FF | Arm CB - BUD Followed by FP | Arm CE - BUD Followed by DISKUS Placebo | Arm DA - ELLIPTA Placebo Followed by FF | EB - DISKUS Placebo Followed by FP | Arm DC - ELLIPTA Placebo Followed by BUD | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD) | ELLIPTA | DISKUS | Total
Number analyzed (Participants) | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 2 | 2 | 3 | 2 | 2 | 7 | 7 | 6 | 3 | 3 | 54
Age, Customized [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
  18 to 64 years | 2 | 3 | 2 | 2 | 3 | 3 | 2 | 2 | 1 | 2 | 2 | 2 | 7 | 7 | 5 | 3 | 2 | 50
  65 to 84 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 13
  Male | 2 | 2 | 1 | 2 | 3 | 2 | 2 | 0 | 1 | 2 | 2 | 2 | 5 | 4 | 5 | 3 | 3 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ASIAN - CENTRAL/SOUTH ASIAN HERITAGE | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4
  ASIAN - EAST ASIAN HERITAGE | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  AFRICAN AMERICAN/AFRICAN HERITAGE | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 7
  WHITE - ARABIC/NORTH AFRICAN HERITAGE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  MULTIPLE | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  WHITE - WHITE/CAUCASIAN/EUROPEAN HERITAGE | 0 | 3 | 1 | 2 | 3 | 1 | 1 | 1 | 1 | 3 | 2 | 2 | 5 | 6 | 4 | 2 | 2 | 39

OUTCOME MEASURES:

1. Primary Outcome: Provocative Concentration (PC) of Adenosine 5' Monophosphate (AMP) Causing a 20 Percent (%) Reduction in Forced Expiratory Volume in 1 Second (FEV1) (AMP PC20)- Dose Response Analysis
Description: The percentage fall in FEV1 was calculated using highest FEV1 (post saline) minus highest FEV1 (post AMP) divided by highest FEV1 (post saline)*100 where highest FEV1 (post saline) is the highest value of two FEV1 measurements at 60 and 180 seconds after the saline control, highest FEV1 (post AMP) is the highest value of the two FEV1 measurements at 60 and 180 seconds after the dose of AMP. Results are presented treatment wise. The analysis method was a 3 parameter Emax model with log 2 transformed AMP PC20 as the outcome variable, assuming common Emax across FF, FP and BUD, and with an unstructured variance-covariance matrix. Mean and 95% Confidence Interval (CI) presented are predicted estimate.
Time Frame: 12 hours post last dose on Day 7
Population: Pharmacodymanic (PD) population. Participants who were randomized and received at least one dose of trial medication and also have at least one post dose PD measurement. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (95% Confidence Interval); unit: Milligrams per milliliter
Groups:
- FF 25 mcg: Participants received placebo FF ELLIPTA 25 mcg 1 puff as total daily dose for 7 days.
- FF 100 mcg: Participants received FF ELLIPTA 100 mcg 1 puff PM as total daily dose for 7 days.
- FF 200 mcg: Participants received FF ELLIPTA 200 mcg 1 puff PM as total daily dose for 7 days.
- FF 400 mcg: Participants received FF ELLIPTA 200 mcg 2 puffs PM as total daily dose for 7 days.
- FF 800 mcg: Participants received FF ELLIPTA 200 mcg 4 puffs PM as total daily dose for 7 days.
- FP 50 mcg: Participants received FF DISKUS 50 mcg 1 puff PM as total daily dose for 7 days.
- FP 200 mcg: Participants received FF DISKUS 100 mcg 1 puff AM and 1 puff PM as total daily dose for 7 days.
- FP 500 mcg: Participants received FF DISKUS 250mcg 1 puff AM and 1 puff PM as total daily dose for 7 days.
- FP 1000 mcg: Participants received FF DISKUS 500 mcg 1 puff AM and 1 puff PM as total daily dose for 7 days.
- FP 2000 mcg: Participants received FF DISKUS 500 mcg 2 puff AM and 2 puff PM as total daily dose for 7 days.
- BUD 100 mcg: Participants received BUD Turbuhaler 100 mcg 1 puff PM as total daily dose for 7 days.
- BUD 400 mcg: Participants received BUD Turbuhaler 200 mcg 1 puff AM and 1 puff PM as total daily dose for 7 days.
- BUD 800 mcg: Participants received BUD Turbuhaler 400 mcg 1 puff AM and 1 puff PM as total daily dose for 7 days.
- BUD 1600 mcg: Participants received BUD Turbuhaler 400 mcg 2 puff AM and 2 puff PM as total daily dose for 7 days.
- BUD 3200 mcg: Participants received BUD Turbuhaler 400 mcg 4 puffs AM and PM as total daily dose for 7 days.
Arm/Group | FF 25 mcg | FF 100 mcg | FF 200 mcg | FF 400 mcg | FF 800 mcg | FP 50 mcg | FP 200 mcg | FP 500 mcg | FP 1000 mcg | FP 2000 mcg | BUD 100 mcg | BUD 400 mcg | BUD 800 mcg | BUD 1600 mcg | BUD 3200 mcg
Number analyzed (Participants) | 19 | 19 | 18 | 18 | 17 | 20 | 20 | 18 | 16 | 17 | 18 | 18 | 18 | 18 | 17
Milligrams per milliliter | 33.45 [19.10 to 58.60] | 81.45 [44.65 to 148.58] | 115.69 [66.82 to 200.31] | 145.97 [85.02 to 250.59] | 167.26 [95.36 to 293.37] | 15.19 [10.80 to 21.36] | 20.47 [13.94 to 30.07] | 31.39 [18.88 to 52.19] | 48.67 [27.30 to 86.78] | 76.35 [43.21 to 134.91] | 16.00 [11.41 to 22.44] | 23.91 [15.08 to 37.90] | 34.62 [19.28 to 62.16] | 54.33 [28.40 to 103.93] | 84.17 [45.48 to 155.79]
Statistical Analysis 1: Comparison: FF 25 mcg vs FF 200 mcg vs FF 400 mcg vs FF 800 mcg; Test type: Other; 3 parameter Emax model = 13.50, 95% CI 2-sided [9.39 to 19.39] — FF E0 (Response of Placebo participants)
Statistical Analysis 2: Comparison: FF 25 mcg vs FF 200 mcg vs FF 400 mcg vs FF 800 mcg; Test type: Other; 3 parameter Emax model = 14.44, 95% CI 2-sided [8.21 to 25.40] — Emax-Maximum Dose response
Statistical Analysis 3: Comparison: FF 25 mcg vs FF 200 mcg vs FF 400 mcg vs FF 800 mcg; Test type: Other; 3 parameter Emax model = 48.52, 95% CI 2-sided [18.21 to 129.32] — ED50-Dose at which 50% of the maximum dose response reached (mcg)
Statistical Analysis 4: Comparison: FP 50 mcg vs FP 200 mcg vs FP 500 mcg vs FP 1000 mcg vs FP 2000 mcg; Test type: Other; 3 parameter Emax model = 13.50, 95% CI 2-sided [9.39 to 19.39] — FP E0-Response of Placebo participants
Statistical Analysis 5: Comparison: FP 50 mcg vs FP 200 mcg vs FP 500 mcg vs FP 1000 mcg vs FP 2000 mcg; Test type: Other; 3 parameter Emax model = 14.44, 95% CI 2-sided [8.21 to 25.40] — FP Emax-Maximum Dose response
Statistical Analysis 6: Comparison: FP 50 mcg vs FP 200 mcg vs FP 500 mcg vs FP 1000 mcg vs FP 2000 mcg; Test type: Other; 3 parameter Emax model = 1081.27, 95% CI 2-sided [448.00 to 2609.66] — FP ED50-Dose at which 50% of the maximum dose response reached (mcg)
Statistical Analysis 7: Comparison: BUD 100 mcg vs BUD 400 mcg vs BUD 800 mcg vs BUD 1600 mcg vs BUD 3200 mcg; Test type: Other; 3 parameter Emax model = 13.50, 95% CI 2-sided [9.39 to 19.39] — BUD E0-Response of Placebo participants
Statistical Analysis 8: Comparison: BUD 100 mcg vs BUD 400 mcg vs BUD 800 mcg vs BUD 1600 mcg vs BUD 3200 mcg; Test type: Other; 3 parameter Emax model = 14.44, 95% CI 2-sided [8.21 to 25.40] — BUD Emax-Maximum Dose response
Statistical Analysis 9: Comparison: BUD 100 mcg vs BUD 400 mcg vs BUD 800 mcg vs BUD 1600 mcg vs BUD 3200 mcg; Test type: Other; 3 parameter Emax model = 1467.36, 95% CI 2-sided [546.51 to 3939.84] — BUD ED50-Dose at which 50% of the maximum dose response reached (mcg)

2. Primary Outcome: Cortisol Suppression 0-24 Hours Weighted Mean-Dose Response Analysis
Description: Blood samples for measurement of plasma cortisol were collected at given time point. The weighted means were derived by calculating the area under the curve (AUC) over the 0-24-hour period using the trapezoidal rule, and then dividing it by the actual time interval. Results are presented treatment wise. Mean and 95% CI presented are predicted estimate. The analysis method was an inhibitory exponential power-law model with log e transformed cortisol as the outcome variable, assuming 100% inhibition at highest doses.
Time Frame: Pre-dose PM dose on Day 6 to pre-dose PM dose Day 7
Population: PD population. Only those participants with data available for each dose escalation phase were analyzed.
Measure: Mean (95% Confidence Interval); unit: nanomoles per liter
Arm/Group | FF 25 mcg | FF 100 mcg | FF 200 mcg | FF 400 mcg | FF 800 mcg | FP 50 mcg | FP 200 mcg | FP 500 mcg | FP 1000 mcg | FP 2000 mcg | BUD 100 mcg | BUD 400 mcg | BUD 800 mcg | BUD 1600 mcg | BUD 3200 mcg
Number analyzed (Participants) | 19 | 19 | 18 | 18 | 18 | 20 | 19 | 18 | 16 | 16 | 16 | 16 | 18 | 18 | 17
nanomoles per liter | 172.73 [159.88 to 186.62] | 163.03 [151.01 to 176.02] | 150.95 [139.48 to 163.37] | 129.40 [117.82 to 142.12] | 95.09 [82.26 to 109.93] | 173.04 [160.15 to 186.97] | 164.22 [152.11 to 177.29] | 147.89 [136.59 to 160.13] | 124.21 [112.88 to 136.68] | 87.62 [75.37 to 101.85] | 169.87 [157.23 to 183.52] | 152.50 [141.26 to 164.63] | 132.06 [122.05 to 142.90] | 99.05 [90.24 to 108.72] | 55.71 [48.26 to 64.31]
Statistical Analysis 1: Comparison: FF 25 mcg vs FF 100 mcg vs FF 200 mcg vs FF 400 mcg; Test type: Other; Exponential power-law model = 176.09, 95% CI 2-sided [162.87 to 190.38] — FF E0-Response of Placebo participants
Statistical Analysis 2: Comparison: FF 25 mcg vs FF 100 mcg vs FF 200 mcg vs FF 400 mcg vs FF 800 mcg; Test type: Other; exponential power-law model = 899.99, 95% CI 2-sided [698.36 to 1101.62] — FF ED50 Dose at which 50% of the maximum dose response reached
Statistical Analysis 3: Comparison: FP 50 mcg vs FP 200 mcg vs FP 500 mcg vs FP 1000 mcg vs FP 2000 mcg; Test type: Other; exponential power-law model = 176.09, 95% CI 2-sided [162.87 to 190.38] — FP E0-Response of Placebo participants
Statistical Analysis 4: Comparison: FP 50 mcg vs FP 200 mcg vs FP 500 mcg vs FP 1000 mcg vs FP 2000 mcg; Test type: Other; exponential power-law model = 1986.05, 95% CI 2-sided [1574.70 to 2397.39] — FP ED50 - Dose at which 50% of the maximum dose response reached (mcg)
Statistical Analysis 5: Comparison: BUD 100 mcg vs BUD 400 mcg vs BUD 800 mcg vs BUD 1600 mcg; Test type: Other; exponential power-law model = 176.09, 95% CI 2-sided [162.87 to 190.38] — BUD E0 - Response of Placebo participants
Statistical Analysis 6: Comparison: BUD 100 mcg vs BUD 400 mcg vs BUD 800 mcg vs BUD 1600 mcg vs BUD 3200 mcg; Test type: Other; exponential power-law model = 1927.42, 95% CI 2-sided [1698.47 to 2156.37] — BUD ED50 - Dose at which 50% of the maximum dose response reached (mcg)

3. Primary Outcome: Theraputic Index of FF
Description: Therapeutic Index was calculated by ED20 for Cortisol Suppression 0-24 Hours Weighted Mean (nanomoles per liter[nmol/L]) divided by Dose at which 80% of the maximum effect is reached (ED80) for AMP PC20 for FF 25 mcg, FF 100 mcg, FF 200 mcg, FF 400 mcg, FF 800 mcg. Theraputic index has been presented. Only those participants with data available at the specified time points were analyzed. The timeframe mentioned is for AMP PC20 and Cortisol suppression respectively.
Time Frame: 12 hours post-dose on Day 7, pre-dose PM dose on Day 6 to pre-dose PM dose Day 7
Population: PD population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Ratio
Groups:
- Fluticasone Propionate (FP): Participants received FF ELLIPTA 25 mcg, 100 mcg, 200 mcg, 400 mcg, 800 mcg for 7 days.
Arm/Group | Fluticasone Propionate (FP)
Number analyzed (Participants) | 51
Ratio | 1.49
Statistical Analysis 1: Comparison: Fluticasone Propionate (FP); Test type: Other; Emax Model = 289.73, 95% CI 2-sided [224.82 to 354.64] — ED20 Cortisol Suppression 0-24 Hours Weighted Mean
Statistical Analysis 2: Comparison: Fluticasone Propionate (FP); Test type: Other; Emax Model = 194.09, 95% CI 2-sided [72.82 to 517.28] — ED80 for AMP PC20

4. Primary Outcome: Theraputic Index of FP
Description: Therapeutic Index was calculated by Dose at which 20% of the maximum effect is reached (ED20) for Cortisol Suppression 0-24 Hours Weighted Mean (nanomoles per liter[nmol/L]) divided by ED80 for AMP PC20 for FP 50 mcg, FP 200 mcg, FP 500 mcg, FP 1000 mcg, FP 2000 mcg. Theraputic index has been presented. The timeframe mentioned is for AMP PC20 and Cortisol suppression respectively.
Time Frame: 12 hours post-dose on Day 7, pre-dose PM dose on Day 6 to pre-dose PM dose Day 7
Population: PD population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Ratio
Groups:
- Fluticasone Propionate (FP): Participants received FP ELLIPTA 50 mg, 200 mcg, 500 mcg, 1000 mcg, 2000 mcg for 7 days.
Arm/Group | Fluticasone Propionate (FP)
Number analyzed (Participants) | 51
Ratio | 0.15
Statistical Analysis 1: Comparison: Fluticasone Propionate (FP); Test type: Other; Emax Model = 639.36, 95% CI 2-sided [506.94 to 771.79] — ED20 for Cortisol Suppression 0-24 Hours Weighted Mean
Statistical Analysis 2: Comparison: Fluticasone Propionate (FP); Test type: Other; Emax Model = 4325.07, 95% CI 2-sided [1792.02 to 10438.64] — ED80 for AMP PC20

5. Primary Outcome: Theraputic Index of BUD
Description: Therapeutic Index was calculated by ED20 for Cortisol Suppression 0-24 Hours Weighted Mean (nanomoles per liter[nmol/L]) divided by ED80 for AMP PC20 for BUD 100 mcg, BUD 400 mcg, BUD 800 mcg, BUD 1600 mcg, BUD 3200 mcg. Theraputic index has been presented. The timeframe mentioned is for AMP PC20 and Cortisol suppression respectively.
Time Frame: 12 hours post-dose on Day 7, pre-dose PM dose on Day 6 to pre-dose PM dose Day 7
Population: PD population. Only those participants with data available at the specified time points were analyzed.
Measure: Number; unit: Ratio
Arm/Group | Budesonide (BUD)
Number analyzed (Participants) | 51
Ratio | 0.11
Statistical Analysis 1: Comparison: Budesonide (BUD); Test type: Other; Emax Model = 620.49, 95% CI 2-sided [546.79 to 694.20] — ED20 for Cortisol Suppression 0-24 Hours Weighted Mean
Statistical Analysis 2: Comparison: Budesonide (BUD); Test type: Other; Emax Model = 5869.45, 95% CI 2-sided [2186.03 to 15759.35] — ED80 for AMP PC20

6. Secondary Outcome: Number of Participants With Any Adverse Event (AE) and Any Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is any untoward medical occurrence that at any dose results in death, Is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect. Results are presented treatment wise.
Time Frame: Up to Week 18
Population: All Subjects Population was consisted of all participants who were randomized and who received at least one dose of trial medication.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received matching placebo ELLIPTA or DISKUS as total daily dose for 7 days.
Arm/Group | Placebo | FF 25 mcg | FF 100 mcg | FF 200 mcg | FF 400 mcg | FF 800 mcg | FP 50 mcg | FP 200 mcg | FP 500 mcg | FP 1000 mcg | FP 2000 mcg | BUD 100 mcg | BUD 400 mcg | BUD 800 mcg | BUD 1600 mcg | BUD 3200 mcg
Number analyzed (Participants) | 17 | 20 | 19 | 19 | 18 | 18 | 21 | 20 | 20 | 18 | 17 | 18 | 18 | 18 | 18 | 18
Participants
  Any AEs | 10 | 6 | 8 | 7 | 6 | 7 | 10 | 4 | 4 | 8 | 6 | 6 | 8 | 5 | 6 | 3
  Any SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability of Placebo in Period 1
Description: PEFR is a participant's maximum speed of expiration and was measured using a peak flow meter. Participants recorded their PEFR measurement before each dose in a paper diary. Results are presented treatment wise.Only those participants with data available at the indicated time points were analyzed (represented by n=X in the category titles).
Time Frame: Day 2 to 8 PM, Day 9 to 14 AM and PM, Day 15 PM, Day 16 to 21 AM and PM, Day 22 PM,Day 23 to 28 AM and PM, Day 29 PM,Day 30 to 35 AM and PM in period 1
Population: All subjects Population.
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | Placebo
Number analyzed (Participants) | 12
Liters per minute
  Day 2, PM, n=12 | 522.5 (25.4)
  Day 3, PM, n=12 | 517.5 (27.0)
  Day 4, PM, n=12 | 514.2 (27.8)
  Day 5,PM, n=12 | 521.7 (24.2)
  Day 6, PM, n=12 | 522.5 (29.1)
  Day 7, PM, n=12 | 539.2 (32.3)
  Day 8, PM, n=12 | 530.8 (27.8)
  Day 9, AM, n=5: number analyzed (Participants) | 5
  Day 9, AM, n=5 | 576.0 (37.5)
  Day 9, PM, n=12 | 531.3 (27.9)
  Day 10, AM, n=5: number analyzed (Participants) | 5
  Day 10, AM, n=5 | 572.0 (34.4)
  Day 10, PM, n=12 | 535.0 (22.0)
  Day 11, AM, n=5: number analyzed (Participants) | 5
  Day 11, AM, n=5 | 578.0 (35.9)
  Day 11, PM, n=12 | 533.8 (29.0)
  Day 12, AM, n=5: number analyzed (Participants) | 5
  Day 12, AM, n=5 | 578.0 (37.2)
  Day 12 PM, n=12 | 527.5 (26.7)
  Day 13, AM, n=5: number analyzed (Participants) | 5
  Day 13, AM, n=5 | 580.0 (37.4)
  Day 13, PM, n=12 | 540.8 (25.1)
  Day 14, AM, n=5: number analyzed (Participants) | 5
  Day 14, AM, n=5 | 572.0 (34.7)
  Day 14, PM, n=12 | 543.3 (26.4)
  Day 15, PM, n=12 | 530.8 (26.0)
  Day 16, AM, n=5: number analyzed (Participants) | 5
  Day 16, AM, n=5 | 588.0 (36.1)
  Day 16,PM, n=12 | 528.3 (24.4)
  Day 17, AM, n=5: number analyzed (Participants) | 5
  Day 17, AM, n=5 | 586.0 (31.7)
  Day 17,PM, n=12 | 521.7 (32.5)
  Day 18, AM, n=5: number analyzed (Participants) | 5
  Day 18, AM, n=5 | 586.0 (35.0)
  Day 18,PM, n=12 | 540.0 (26.9)
  Day 19, AM, n=5: number analyzed (Participants) | 5
  Day 19, AM, n=5 | 568.0 (38.3)
  Day 19,PM, n=12 | 535.8 (29.3)
  Day 20, AM, n=5: number analyzed (Participants) | 5
  Day 20, AM, n=5 | 596.0 (37.5)
  Day 20,PM, n=12 | 544.2 (28.2)
  Day 21, AM, n=5: number analyzed (Participants) | 5
  Day 21, AM, n=5 | 580.0 (31.4)
  Day 21,PM, n=12 | 534.2 (32.6)
  Day 22,PM, n=11: number analyzed (Participants) | 11
  Day 22,PM, n=11 | 544.5 (29.0)
  Day 23, AM, n=4: number analyzed (Participants) | 4
  Day 23, AM, n=4 | 577.5 (37.9)
  Day 23,PM, n=11: number analyzed (Participants) | 11
  Day 23,PM, n=11 | 530.0 (27.4)
  Day 24, AM, n=4: number analyzed (Participants) | 4
  Day 24, AM, n=4 | 567.5 (39.4)
  Day 24,PM, n=11: number analyzed (Participants) | 11
  Day 24,PM, n=11 | 526.4 (26.5)
  Day 25, AM, n=4: number analyzed (Participants) | 4
  Day 25, AM, n=4 | 585.0 (39.2)
  Day 25,PM, n=11: number analyzed (Participants) | 11
  Day 25,PM, n=11 | 530.9 (29.6)
  Day 26, AM, n=4: number analyzed (Participants) | 4
  Day 26, AM, n=4 | 582.5 (40.0)
  Day 26,PM, n=11: number analyzed (Participants) | 11
  Day 26,PM, n=11 | 518.2 (30.0)
  Day 27, AM, n=4: number analyzed (Participants) | 4
  Day 27, AM, n=4 | 587.5 (40.0)
  Day 27,PM, n=11: number analyzed (Participants) | 11
  Day 27,PM, n=11 | 539.1 (29.3)
  Day 28, AM, n=4: number analyzed (Participants) | 4
  Day 28, AM, n=4 | 587.5 (43.0)
  Day 28,PM, n=10: number analyzed (Participants) | 10
  Day 28,PM, n=10 | 547.0 (30.4)
  Day 29,PM, n=11: number analyzed (Participants) | 11
  Day 29,PM, n=11 | 547.3 (28.2)
  Day 30, AM, n=4: number analyzed (Participants) | 4
  Day 30, AM, n=4 | 567.5 (38.1)
  Day 30,PM, n=11: number analyzed (Participants) | 11
  Day 30,PM, n=11 | 527.3 (26.6)
  Day 31, AM, n=4: number analyzed (Participants) | 4
  Day 31, AM, n=4 | 562.5 (33.2)
  Day 31,PM, n=11: number analyzed (Participants) | 11
  Day 31,PM, n=11 | 537.3 (26.5)
  Day 32, AM, n=4: number analyzed (Participants) | 4
  Day 32, AM, n=4 | 582.5 (40.2)
  Day 32,PM, n=11: number analyzed (Participants) | 11
  Day 32,PM, n=11 | 537.3 (26.2)
  Day 33, AM, n=4: number analyzed (Participants) | 4
  Day 33, AM, n=4 | 597.5 (40.0)
  Day 33,PM, n=11: number analyzed (Participants) | 11
  Day 33,PM, n=11 | 528.2 (30.5)
  Day 34, AM, n=4: number analyzed (Participants) | 4
  Day 34, AM, n=4 | 580.0 (39.3)
  Day 34,PM, n=11: number analyzed (Participants) | 11
  Day 34,PM, n=11 | 531.4 (31.9)
  Day 35, AM, n=4: number analyzed (Participants) | 4
  Day 35, AM, n=4 | 565.0 (38.8)
  Day 35,PM, n=11: number analyzed (Participants) | 11
  Day 35,PM, n=11 | 501.8 (26.1)

8. Secondary Outcome: PEFR as a Measure of Safety and Tolerability of Placebo in Period 2
Description: PEFR is a participant's maximum speed of expiration and was measured using a peak flow meter. Participants recorded their PEFR measurement before each dose in a paper diary. Results are presented treatment wise.
Time Frame: Day 2 to 8 PM, Day 9 to 14 AM and PM, Day 15 PM, Day 16 to 21 AM and PM, Day 22 PM,Day 23 to 28 AM and PM, Day 29 PM,Day 30 to 35 AM and PM in Period 2
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed (represented by n=X in the category titles).
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | Placebo
Number analyzed (Participants) | 4
Liters per minute
  Day 2, PM, n=4 | 422.5 (28.9)
  Day 3, PM, n=4 | 415.0 (27.2)
  Day 4, PM, n=4 | 398.8 (26.6)
  Day 5,PM, n=4 | 407.5 (37.5)
  Day 6, PM, n=4 | 411.3 (29.0)
  Day 7, PM, n=4 | 410.0 (36.7)
  Day 8, PM, n=4 | 415.0 (36.1)
  Day 9, AM, n=2: number analyzed (Participants) | 2
  Day 9, AM, n=2 | 430.0 (80.0)
  Day 9, PM, n=4 | 411.3 (45.4)
  Day 10, AM, n=2: number analyzed (Participants) | 2
  Day 10, AM, n=2 | 425.0 (65.0)
  Day 10, PM, n=4 | 403.8 (37.1)
  Day 11, AM, n=2: number analyzed (Participants) | 2
  Day 11, AM, n=2 | 410.0 (60.0)
  Day 11, PM, n=4 | 395.0 (29.0)
  Day 12, AM, n=2: number analyzed (Participants) | 2
  Day 12, AM, n=2 | 400.0 (50.0)
  Day 12, PM, n=4 | 398.8 (28.6)
  Day 13, AM, n=2: number analyzed (Participants) | 2
  Day 13, AM, n=2 | 415.0 (95.0)
  Day 13, PM, n=4 | 425.0 (35.2)
  Day 14, AM, n=2: number analyzed (Participants) | 2
  Day 14, AM, n=2 | 425.0 (65.0)
  Day 14, PM, n=3: number analyzed (Participants) | 3
  Day 14, PM, n=3 | 420.0 (40.4)
  Day 15, PM, n=4 | 416.3 (37.0)
  Day 16, AM, n=2: number analyzed (Participants) | 2
  Day 16, AM, n=2 | 405.0 (75.0)
  Day 16,PM, n=4 | 405.0 (32.0)
  Day 17, AM, n=2: number analyzed (Participants) | 2
  Day 17, AM, n=2 | 390.0 (70.0)
  Day 17,PM, n=4 | 405.0 (28.9)
  Day 18, AM, n=1: number analyzed (Participants) | 1
  Day 18, AM, n=1 | 450.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 18,PM,n=3: number analyzed (Participants) | 3
  Day 18,PM,n=3 | 423.3 (34.8)
  Day 19, AM, n=2: number analyzed (Participants) | 2
  Day 19, AM, n=2 | 415.0 (65.0)
  Day 19,PM, n=4 | 402.5 (30.1)
  Day 20, AM, n=2: number analyzed (Participants) | 2
  Day 20, AM, n=2 | 402.5 (57.5)
  Day 20,PM, n=4 | 398.8 (36.3)
  Day 21, AM, n=2: number analyzed (Participants) | 2
  Day 21, AM, n=2 | 400.0 (60.0)
  Day 21,PM, n=4 | 395.0 (38.6)
  Day 22,PM, n=4 | 397.5 (34.9)
  Day 23, AM, n=1: number analyzed (Participants) | 1
  Day 23, AM, n=1 | 480.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 23,PM, n=3: number analyzed (Participants) | 3
  Day 23,PM, n=3 | 415.0 (39.0)
  Day 24, AM, n=1: number analyzed (Participants) | 1
  Day 24, AM, n=1 | 460.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 24,PM, n=3: number analyzed (Participants) | 3
  Day 24,PM, n=3 | 423.3 (38.4)
  Day 25, AM, n=1: number analyzed (Participants) | 1
  Day 25, AM, n=1 | 460.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 25,PM, n=3: number analyzed (Participants) | 3
  Day 25,PM, n=3 | 416.7 (33.8)
  Day 26, AM, n=1: number analyzed (Participants) | 1
  Day 26, AM, n=1 | 450.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 26,PM, n=3: number analyzed (Participants) | 3
  Day 26,PM, n=3 | 418.3 (36.7)
  Day 27, AM, n=1: number analyzed (Participants) | 1
  Day 27, AM, n=1 | 460.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 27,PM, n=3: number analyzed (Participants) | 3
  Day 27,PM, n=3 | 433.3 (49.7)
  Day 28, AM, n=1: number analyzed (Participants) | 1
  Day 28, AM, n=1 | 460.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 28,PM, n=3: number analyzed (Participants) | 3
  Day 28,PM, n=3 | 430.0 (49.3)
  Day 29,PM, n=3: number analyzed (Participants) | 3
  Day 29,PM, n=3 | 380.0 (75.5)
  Day 30, AM, n=1: number analyzed (Participants) | 1
  Day 30, AM, n=1 | 460.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 30,PM, n=3: number analyzed (Participants) | 3
  Day 30,PM, n=3 | 388.3 (78.0)
  Day 31, AM, n=1: number analyzed (Participants) | 1
  Day 31, AM, n=1 | 480.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 31,PM, n=3: number analyzed (Participants) | 3
  Day 31,PM, n=3 | 390.0 (85.0)
  Day 32, AM, n=1: number analyzed (Participants) | 1
  Day 32, AM, n=1 | 500.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 32,PM, n=3: number analyzed (Participants) | 3
  Day 32,PM, n=3 | 370.0 (73.7)
  Day 33, AM, n=1: number analyzed (Participants) | 1
  Day 33, AM, n=1 | 470.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 33,PM, n=3: number analyzed (Participants) | 3
  Day 33,PM, n=3 | 370.0 (70.9)
  Day 34, AM, n=1: number analyzed (Participants) | 1
  Day 34, AM, n=1 | 460.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 34,PM, n=3: number analyzed (Participants) | 3
  Day 34,PM, n=3 | 390.0 (83.2)
  Day 35, AM, n=1: number analyzed (Participants) | 1
  Day 35, AM, n=1 | 480.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 35,PM, n=2: number analyzed (Participants) | 2
  Day 35,PM, n=2 | 345.0 (105.0)

9. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FF 25 mcg in Period 1
Description: PEFR is a participant's maximum speed of expiration and was measured using a peak flow meter. Results are presented treatment wise.
Time Frame: Day 2,3,4,5,6,7 PM in period 1
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Error); unit: Liters per minute
Groups:
- FF 25 mcg: Participants received FF ELLIPTA 25 mcg 1 puff PM as total daily dose for 7 days
Arm/Group | FF 25 mcg
Number analyzed (Participants) | 14
Liters per minute
  Day 2, PM, n=14 | 479.6 (30.9)
  Day 3, PM, n=14 | 475.7 (32.9)
  Day 4, PM, n=14 | 473.0 (31.1)
  Day 5,PM, n=14 | 476.1 (26.6)
  Day 6, PM, n=13: number analyzed (Participants) | 13
  Day 6, PM, n=13 | 503.1 (24.6)
  Day 7, PM, n=13: number analyzed (Participants) | 13
  Day 7, PM, n=13 | 502.3 (28.1)

10. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FF 25 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 2,3,4,5,6,7 PM in period 2
Population: as for outcome 9
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | FF 25 mcg
Number analyzed (Participants) | 6
Liters per minute
  Day 2, PM, n=5: number analyzed (Participants) | 5
  Day 2, PM, n=5 | 572.0 (48.9)
  Day 3, PM, n=5: number analyzed (Participants) | 5
  Day 3, PM, n=5 | 570.0 (54.5)
  Day 4, PM, n=5: number analyzed (Participants) | 5
  Day 4, PM, n=5 | 568.0 (55.0)
  Day 5,PM, n=5: number analyzed (Participants) | 5
  Day 5,PM, n=5 | 573.0 (54.9)
  Day 6, PM, n=6 | 550.8 (52.2)
  Day 7, PM, n=6 | 560.0 (45.3)

11. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FF 100 mcg in Period 1
Description: as for outcome 9
Time Frame: Day 8,9,10,11,12,13,14 PM in period 1
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | FF 100 mcg
Number analyzed (Participants) | 13
Liters per minute
  Day 8, PM, n=13 | 497.3 (24.9)
  Day 9, PM, n=13 | 500.4 (28.2)
  Day 10, PM, n=13 | 491.2 (31.0)
  Day 11, PM, n=12: number analyzed (Participants) | 12
  Day 11, PM, n=12 | 507.5 (30.9)
  Day 12, PM, n=13 | 500.2 (30.2)
  Day 13, PM, n=13 | 515.4 (29.7)
  Day 14, PM, n=13 | 505.8 (28.7)

12. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FF 100 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 8,9,10,11,12,13,14 PM in period 2
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | FF 100 mcg
Number analyzed (Participants) | 6
Liters per minute
  Day 8, PM | 540.0 (43.8)
  Day 9, PM | 567.5 (42.6)
  Day 10, PM | 556.7 (43.4)
  Day 11, PM | 561.7 (44.6)
  Day 12, PM | 573.3 (50.0)
  Day 13, PM | 563.3 (53.0)
  Day 14, PM | 555.8 (46.9)

13. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FF 200 mcg in Period 1
Description: as for outcome 9
Time Frame: Day 15,16,17,18,19,20,21 PM in period 1
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | FF 200 mcg
Number analyzed (Participants) | 13
Liters per minute
  Day 15,PM, n=13 | 500.8 (30.8)
  Day 16,PM, n=13 | 500.0 (28.7)
  Day 17,PM, n=13 | 506.2 (29.8)
  Day 18,PM, n=13 | 514.2 (31.6)
  Day 19,PM, n=13 | 505.4 (29.0)
  Day 20,PM, n=12: number analyzed (Participants) | 12
  Day 20,PM, n=12 | 505.8 (30.8)
  Day 21,PM, n=12: number analyzed (Participants) | 12
  Day 21,PM, n=12 | 485.0 (28.2)

14. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FF 200 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 15,16,17,18,19,20 PM, Day 21 AM and PM in period 2
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | FF 200 mcg
Number analyzed (Participants) | 6
Liters per minute
  Day 15,PM, n=6 | 575.0 (52.9)
  Day 16,PM, n=6 | 575.0 (48.1)
  Day 17,PM, n=6 | 564.2 (46.6)
  Day 18,PM, n=6 | 573.3 (56.6)
  Day 19,PM, n=6 | 556.7 (53.4)
  Day 20,PM, n=6 | 571.7 (50.0)
  Day 21,AM, n=1: number analyzed (Participants) | 1
  Day 21,AM, n=1 | 670.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 21,PM, n=6 | 560.0 (38.3)

15. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FF 400 mcg in Period 1
Description: as for outcome 9
Time Frame: Days 22,23,24,25,26,27,28 PM in period 1
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Liters per minute
Groups:
- FF 400 mcg: Participants received FF ELLIPTA 200 mcg 2 puff PM as total daily dose for 7 days
Arm/Group | FF 400 mcg
Number analyzed (Participants) | 12
Liters per minute
  Day 22 PM | 496.7 (30.5)
  Day 23 PM | 481.0 (25.6)
  Day 24 PM | 484.6 (25.2)
  Day 25 PM | 488.3 (26.2)
  Day 26 PM | 496.7 (28.8)
  Day 27 PM | 508.8 (28.9)
  Day 28 PM | 486.7 (23.7)

16. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FF 400 mcg in Period 2
Description: as for outcome 9
Time Frame: Days 22,23,24,25,26,27,28 PM in period 2
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | FF 400 mcg
Number analyzed (Participants) | 6
Liters per minute
  Day 22 PM | 556.7 (46.9)
  Day 23 PM | 566.7 (47.8)
  Day 24 PM | 571.7 (50.8)
  Day 25 PM | 568.3 (52.7)
  Day 26 PM | 565.0 (43.0)
  Day 27 PM | 540.0 (43.3)
  Day 28 PM | 541.7 (41.2)

17. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FF 800 mcg in Period 1
Description: as for outcome 9
Time Frame: Days 29,30,31,32,33,34,35 PM in period 1
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Liters per minute
Groups:
- FF 800 mcg: Participants received FF ELLIPTA 200 mcg 4 puff PM as total daily dose for 7 days
Arm/Group | FF 800 mcg
Number analyzed (Participants) | 12
Liters per minute
  Day 29 PM | 496.7 (27.0)
  Day 30 PM | 487.1 (25.9)
  Day 31 PM | 488.3 (24.1)
  Day 32 PM | 481.3 (25.8)
  Day 33 PM | 481.5 (24.9)
  Day 34 PM | 487.5 (28.7)
  Day 35 PM | 471.0 (26.6)

18. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FF 800 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 29,30,31,32,33,34,35 PM in period 2
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Liters per minute
Groups:
- FF 400 mcg: Participants received FF ELLIPTA 400 mcg 1 puff PM as total daily dose for 7 days
Arm/Group | FF 400 mcg
Number analyzed (Participants) | 6
Liters per minute
  Day 29 PM | 576.7 (44.9)
  Day 30 PM | 560.0 (48.7)
  Day 31 PM | 553.3 (45.0)
  Day 32 PM | 565.0 (50.7)
  Day 33 PM | 580.0 (48.9)
  Day 34 PM | 568.3 (42.3)
  Day 35 PM | 556.7 (44.9)

19. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FP 50 mcg in Period 1
Description: as for outcome 9
Time Frame: Day 2,3,4,5,6,7 PM in period 1
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Groups:
- FP 50 mcg: Participants received FP ELLIPTA 50 mcg 1 puff PM as total daily dose for 7 days
Arm/Group | FP 50 mcg
Number analyzed (Participants) | 15
Liters per minute
  Day 2 PM, n=15 | 529.3 (28.0)
  Day 3 PM, n=14: number analyzed (Participants) | 14
  Day 3 PM, n=14 | 533.6 (30.3)
  Day 4 PM, n=15 | 532.3 (30.8)
  Day 5 PM, n=15 | 524.0 (29.9)
  Day 6 PM, n=14: number analyzed (Participants) | 14
  Day 6 PM, n=14 | 519.3 (26.4)
  Day 7 PM, n=14: number analyzed (Participants) | 14
  Day 7 PM, n=14 | 502.9 (35.1)

20. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FP 50 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 2,3,4,5,6,7 AM and PM in period 2
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | FP 50 mcg
Number analyzed (Participants) | 6
Liters per minute
  Day 2 AM, n=1: number analyzed (Participants) | 1
  Day 2 AM, n=1 | 600.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 2 PM, n=6 | 490.0 (40.6)
  Day 3 AM, n=1: number analyzed (Participants) | 1
  Day 3 AM, n=1 | 600.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 3 PM, n=6 | 486.7 (42.3)
  Day 4 PM, n=1: number analyzed (Participants) | 1
  Day 4 PM, n=1 | 590.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 4 PM, n=6 | 491.7 (42.6)
  Day 5 AM, n=1: number analyzed (Participants) | 1
  Day 5 AM, n=1 | 600.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 5 PM, n=6 | 491.7 (44.6)
  Day 6 PM, n=1: number analyzed (Participants) | 1
  Day 6 PM, n=1 | 600.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 6 PM, n=6 | 490.0 (44.3)
  Day 7 PM, n=1: number analyzed (Participants) | 1
  Day 7 PM, n=1 | 600.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 7 PM, n=6 | 466.0 (48.9)

21. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FP 200 mcg in Period 1
Description: as for outcome 9
Time Frame: Days 8,9,1,0,11,12,13,14 AM and PM in period 1
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Groups:
- FP 200 mcg: Participants received FP DISKSU 200 mcg 1 puff AM and 1 puff PM as total daily dose for 7 days
Arm/Group | FP 200 mcg
Number analyzed (Participants) | 14
Liters per minute
  Day 8 AM, n=1: number analyzed (Participants) | 1
  Day 8 AM, n=1 | 540.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 8 PM, n=13: number analyzed (Participants) | 13
  Day 8 PM, n=13 | 532.7 (33.2)
  Day 9 AM, n=11: number analyzed (Participants) | 11
  Day 9 AM, n=11 | 500.9 (38.3)
  Day 9 PM, n=14 | 517.9 (26.8)
  Day 10 AM, n=10: number analyzed (Participants) | 10
  Day 10 AM, n=10 | 521.0 (39.0)
  Day 10 PM, n=14 | 513.2 (28.5)
  Day 11 AM, n=11: number analyzed (Participants) | 11
  Day 11 AM, n=11 | 476.4 (35.4)
  Day 11 PM, n=14 | 512.1 (30.0)
  Day 12 AM, n=11: number analyzed (Participants) | 11
  Day 12 AM, n=11 | 506.8 (38.0)
  Day 12 PM, n=13: number analyzed (Participants) | 13
  Day 12 PM, n=13 | 528.8 (34.3)
  Day 13 AM, n=11: number analyzed (Participants) | 11
  Day 13 AM, n=11 | 500.0 (38.2)
  Day 13 PM, n=14 | 514.6 (31.1)
  Day 14 AM, n=13: number analyzed (Participants) | 13
  Day 14 AM, n=13 | 496.2 (31.7)
  Day14 PM, n=13: number analyzed (Participants) | 13
  Day14 PM, n=13 | 522.7 (32.9)

22. Secondary Outcome: PEFR as a Measure of Safety and Tolerability for FP 200 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 8,9,1,0,11,12,13,14 AM and PM in period 2
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Groups:
- FP 200 mcg: Participants received FP DISKSUS 100 mcg 1 puff AM and 1 puff PM as total daily dose for 7 days
Arm/Group | FP 200 mcg
Number analyzed (Participants) | 6
Liters per minute
  Day 8 AM, n=1: number analyzed (Participants) | 1
  Day 8 AM, n=1 | 610.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 8 PM, n=6 | 500.0 (43.2)
  Day 9 AM, n=5: number analyzed (Participants) | 5
  Day 9 AM, n=5 | 506.0 (39.5)
  Day 9 PM, n=6 | 488.3 (43.7)
  Day 10 AM, n=4: number analyzed (Participants) | 4
  Day 10 AM, n=4 | 515.0 (44.0)
  Day 10 PM, n=6 | 490.0 (47.1)
  Day 11 AM, n=5: number analyzed (Participants) | 5
  Day 11 AM, n=5 | 504.0 (36.1)
  Day 11 PM, n=6 | 485.0 (42.6)
  Day 12 AM, n=5: number analyzed (Participants) | 5
  Day 12 AM, n=5 | 508.0 (41.4)
  Day 12 PM, n=6 | 493.3 (42.8)
  Day 13 AM, n=5: number analyzed (Participants) | 5
  Day 13 AM, n=5 | 500.0 (40.1)
  Day 13 PM, n=6 | 495.0 (45.8)
  Day 14 AM, n=5: number analyzed (Participants) | 5
  Day 14 AM, n=5 | 438.0 (46.6)
  Day 14 PM, n=6 | 495.8 (48.8)

23. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for FP 500 mcg in Period 1
Description: PEFR is a participant's maximum speed of expiration and was measured using a peak flow meter. Results are presented treatment wise. One participant who was supposed to receive FP 1000 mg during day 22-28 and FP 2000 mg during day 28-35 but this participant continued the 3rd escalation phase dose (FP 500 mg) in fourth escalation phase and took FP 1000 mg (4th phase dose) in the fifth escalation phase (days 28-35).
Time Frame: Day 15 PM, Day 16,17,18,19,20,21,22,23,24,25,26,27,28 AM and PM in period 1
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Groups:
- FP 500 mcg: Participants received FP DISKSUS 250 mcg 1 puff AM and 1 puff PM as total daily dose for 7 days
Arm/Group | FP 500 mcg
Number analyzed (Participants) | 14
Liters per minute
  Day 15 PM, n=14 | 527.5 (29.7)
  Day 16 AM, n=13: number analyzed (Participants) | 13
  Day 16 AM, n=13 | 503.8 (31.9)
  Day 16 PM, n=14 | 520.4 (29.5)
  Day 17 AM, n=13: number analyzed (Participants) | 13
  Day 17 AM, n=13 | 510.0 (30.3)
  Day 17 PM, n=14 | 508.6 (31.2)
  Day 18 AM, n=12: number analyzed (Participants) | 12
  Day 18 AM, n=12 | 497.5 (34.7)
  Day 18 PM, n=13: number analyzed (Participants) | 13
  Day 18 PM, n=13 | 505.8 (28.5)
  Day 19 AM, n=12: number analyzed (Participants) | 12
  Day 19 AM, n=12 | 505.8 (35.2)
  Day 19 PM, n=13: number analyzed (Participants) | 13
  Day 19 PM, n=13 | 506.9 (29.5)
  Day 20 AM, n=11: number analyzed (Participants) | 11
  Day 20 AM, n=11 | 518.2 (35.9)
  Day 20 PM, n=13: number analyzed (Participants) | 13
  Day 20 PM, n=13 | 517.3 (30.4)
  Day 21 AM, n=13: number analyzed (Participants) | 13
  Day 21 AM, n=13 | 501.9 (32.1)
  Day 21 PM, n=11: number analyzed (Participants) | 11
  Day 21 PM, n=11 | 493.6 (30.0)
  Day 22 AM, n=1: number analyzed (Participants) | 1
  Day 22 AM, n=1 | 520.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 22 PM, n=1: number analyzed (Participants) | 1
  Day 22 PM, n=1 | 540.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 23 AM, n=1: number analyzed (Participants) | 1
  Day 23 AM, n=1 | 530.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 23 PM, n=1: number analyzed (Participants) | 1
  Day 23 PM, n=1 | 550.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 24 AM, n=1: number analyzed (Participants) | 1
  Day 24 AM, n=1 | 530.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 24 PM, n=1: number analyzed (Participants) | 1
  Day 24 PM, n=1 | 540.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 25 AM, n=1: number analyzed (Participants) | 1
  Day 25 AM, n=1 | 510.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 25 PM, n=1: number analyzed (Participants) | 1
  Day 25 PM, n=1 | 500.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 26 AM, n=1: number analyzed (Participants) | 1
  Day 26 AM, n=1 | 520.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 26 PM, n=1: number analyzed (Participants) | 1
  Day 26 PM, n=1 | 550.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 27 AM, n=1: number analyzed (Participants) | 1
  Day 27 AM, n=1 | 530.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 27 PM, n=1: number analyzed (Participants) | 1
  Day 27 PM, n=1 | 580.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 28 AM, n=1: number analyzed (Participants) | 1
  Day 28 AM, n=1 | 530.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 28 PM, n=1: number analyzed (Participants) | 1
  Day 28 PM, n=1 | 500.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.

24. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for FP 500 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 15 PM, Day 16,17,18,19,20,21 AM and PM in period 2
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Groups:
- FP 500 mcg: Participants received FP DISKUS 250 mcg 1 puff AM and 1 puff PM as total daily dose for 7 days
Arm/Group | FP 500 mcg
Number analyzed (Participants) | 6
Liters per minute
  Day 15 PM, n=6 | 486.7 (43.8)
  Day 16 AM, n=6 | 476.7 (43.8)
  Day 16 PM, n=6 | 503.3 (46.8)
  Day 17 AM, n=6 | 493.3 (44.0)
  Day 17 PM, n=6 | 500.0 (45.9)
  Day 18 AM, n=6 | 476.7 (39.9)
  Day 18 PM, n=6 | 495.0 (42.8)
  Day 19 AM, n=5: number analyzed (Participants) | 5
  Day 19 AM, n=5 | 454.0 (44.3)
  Day 19 PM, n=6 | 500.0 (45.1)
  Day 20 AM, n=5: number analyzed (Participants) | 5
  Day 20 AM, n=5 | 524.0 (43.6)
  Day 20 PM, n=6 | 501.7 (50.6)
  Day 21 AM, n=6 | 490.0 (44.2)
  Day 21 PM, n=6 | 496.7 (48.4)

25. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for FP 1000 mcg in Period 1
Description: as for outcome 23
Time Frame: Day 22 PM, Day 23,24,25,26,27,28,29,30,31,32,33,34,35 AM and PM in period 1
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Groups:
- FP 1000 mcg: Participants received FP DISKSUS 500 mcg 1 puff AM and 1 puff PM as total daily dose for 7 days
Arm/Group | FP 1000 mcg
Number analyzed (Participants) | 11
Liters per minute
  Day 22 PM, n=6: number analyzed (Participants) | 6
  Day 22 PM, n=6 | 523.2 (30.5)
  Day 23 AM, n=11 | 511.8 (36.4)
  Day 23 PM, n=11 | 516.4 (38.4)
  Day 24 AM, n=11 | 521.8 (38.0)
  Day 24 PM, n=11 | 520.9 (37.1)
  Day 25 AM, n=11 | 489.5 (35.1)
  Day 25 PM, n=10: number analyzed (Participants) | 10
  Day 25 PM, n=10 | 521.0 (42.7)
  Day 26 AM, n=11 | 502.7 (37.0)
  Day 26 PM, n=11 | 517.3 (35.7)
  Day 27 AM, n=11 | 493.6 (33.0)
  Day 27 PM, n=11 | 523.6 (37.7)
  Day 28 AM, n=11 | 500.0 (40.6)
  Day 28,PM, n=11 | 516.4 (33.9)
  Day 29 PM, n=1: number analyzed (Participants) | 1
  Day 29 PM, n=1 | 530.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 30 AM, n=1: number analyzed (Participants) | 1
  Day 30 AM, n=1 | 520.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed..
  Day 30 PM, n=1: number analyzed (Participants) | 1
  Day 30 PM, n=1 | 530.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 31 AM, n=1: number analyzed (Participants) | 1
  Day 31 AM, n=1 | 510.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 31 PM, n=1: number analyzed (Participants) | 1
  Day 31 PM, n=1 | 530.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 32 AM, n=1: number analyzed (Participants) | 1
  Day 32 AM, n=1 | 520.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 32 PM, n=1: number analyzed (Participants) | 1
  Day 32 PM, n=1 | 550.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 33 AM, n=1: number analyzed (Participants) | 1
  Day 33 AM, n=1 | 530.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 33 PM, n=1: number analyzed (Participants) | 1
  Day 33 PM, n=1 | 540.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 34 AM, n=1: number analyzed (Participants) | 1
  Day 34 AM, n=1 | 510.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 34 PM, n=1: number analyzed (Participants) | 1
  Day 34 PM, n=1 | 520.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 35 AM, n=1: number analyzed (Participants) | 1
  Day 35 AM, n=1 | 540.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 35 PM, n=1: number analyzed (Participants) | 1
  Day 35 PM, n=1 | 550.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.

26. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for FP 1000 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 22 PM, Day 23,24,25,26,27,28 AM and PM in period 2
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | FP 1000 mcg
Number analyzed (Participants) | 6
Liters per minute
  Day 22 PM, n=6 | 493.3 (42.8)
  Day 23 AM, n=6 | 480.0 (43.4)
  Day 23 PM, n=6 | 506.7 (43.5)
  Day 24 AM, n=6 | 481.7 (39.4)
  Day 24 PM, n=6 | 505.0 (45.3)
  Day 25 AM, n=6 | 491.7 (43.9)
  Day 25 PM, n=6 | 510.0 (51.7)
  Day 26 AM, n=6 | 485.0 (45.3)
  Day 26 PM, n=6 | 501.7 (49.9)
  Day 27 AM, n=6 | 475.0 (42.3)
  Day 27 PM, n=6 | 490.0 (43.2)
  Day 28 AM, n=5: number analyzed (Participants) | 5
  Day 28 AM, n=5 | 452.0 (47.7)
  Day 28,PM, n=5: number analyzed (Participants) | 5
  Day 28,PM, n=5 | 476.0 (56.8)

27. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for FP 2000 mcg in Period 1
Description: as for outcome 9
Time Frame: Day 29 PM, Day 30,31,32,33,34,35 AM and PM in period 1
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Groups:
- FP 2000 mcg: Participants received FP DISKSU 500 mcg 2 puffs AM and 2 puffs PM as total daily dose for 7 days.
Arm/Group | FP 2000 mcg
Number analyzed (Participants) | 10
Liters per minute
  Day 29 PM, n=10 | 520.5 (36.5)
  Day 30 AM, n=10 | 505.0 (39.0)
  Day 30 PM, n=10 | 520.0 (40.9)
  Day 31 AM, n=10 | 507.0 (37.0)
  Day 31 PM, n=10 | 521.0 (41.7)
  Day 32 AM, n=10 | 500.0 (39.6)
  Day 32 PM, n=10 | 524.0 (41.9)
  Day 33 AM, n=10 | 511.0 (40.7)
  Day 33 PM, n=10 | 511.5 (43.2)
  Day 34 AM, n=10 | 519.0 (38.9)
  Day 34 PM, n=10 | 517.0 (38.9)
  Day 35 AM, n=9: number analyzed (Participants) | 9
  Day 35 AM, n=9 | 514.4 (40.4)
  Day 35 PM, n=9: number analyzed (Participants) | 9
  Day 35 PM, n=9 | 543.9 (44.1)

28. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for FP 2000 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 29 PM, Day 30,31,32,33,34,35 AM and PM in period 2
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | FP 2000 mcg
Number analyzed (Participants) | 6
Liters per minute
  Day 29 PM | 506.7 (45.8)
  Day 30 AM | 493.3 (45.0)
  Day 30 PM | 496.7 (46.8)
  Day 31 AM | 486.7 (48.0)
  Day 31 PM | 485.0 (41.6)
  Day 32 AM | 488.3 (44.7)
  Day 32 PM | 513.3 (52.6)
  Day 33 AM | 495.0 (45.3)
  Day 33 PM | 498.3 (44.1)
  Day 34 AM | 481.7 (46.0)
  Day 34 PM | 498.3 (47.7)
  Day 35 AM | 483.3 (44.2)
  Day 35 PM | 493.3 (46.3)

29. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for BUD 100 mcg in Period 1
Description: as for outcome 9
Time Frame: Day 2 to 6 AM and PM, Day 7 PM in period 1
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | BUD 100 mcg
Number analyzed (Participants) | 12
Liters per minute
  Day 2 AM, n=1: number analyzed (Participants) | 1
  Day 2 AM, n=1 | 600.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 2 PM, n=12 | 512.9 (33.4)
  Day 3 AM, n=1: number analyzed (Participants) | 1
  Day 3 AM, n=1 | 600.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 3 PM, n=12 | 517.1 (31.2)
  Day 4 AM, n=1: number analyzed (Participants) | 1
  Day 4 AM, n=1 | 625.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 4 PM, n=12 | 524.2 (32.9)
  Day 5 AM, n=1: number analyzed (Participants) | 1
  Day 5 AM, n=1 | 600.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 5 PM, n=12 | 520.8 (32.3)
  Day 6 AM, n=1: number analyzed (Participants) | 1
  Day 6 AM, n=1 | 600.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 6 PM, n=12 | 523.3 (33.5)
  Day 7 PM, n=12 | 527.5 (33.4)

30. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for BUD 100 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 2,3,4,5,6,7 PM in period 2
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | BUD 100 mcg
Number analyzed (Participants) | 4
Liters per minute
  Day 2 PM, n=4 | 557.5 (28.3)
  Day 3 PM, n=4 | 547.5 (60.1)
  Day 4 PM, n=4 | 545.0 (27.2)
  Day 5 PM, n=4 | 552.5 (46.0)
  Day 6 PM, n=4 | 577.5 (26.5)
  Day 7 PM, n=3: number analyzed (Participants) | 3
  Day 7 PM, n=3 | 603.3 (32.8)

31. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for BUD 400 mcg in Period 1
Description: as for outcome 9
Time Frame: Day 8 PM, Day 9 to 14 AM and PM in period 1
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | BUD 400 mcg
Number analyzed (Participants) | 12
Liters per minute
  Day 8 PM, n=12 | 521.7 (31.5)
  Day 9 AM, n=10: number analyzed (Participants) | 10
  Day 9 AM, n=10 | 473.0 (30.5)
  Day 9 PM, n=12 | 515.4 (34.3)
  Day 10 AM, n=10: number analyzed (Participants) | 10
  Day 10 AM, n=10 | 470.0 (33.9)
  Day 10 PM, n=12 | 512.9 (32.8)
  Day 11 AM, n=10: number analyzed (Participants) | 10
  Day 11 AM, n=10 | 466.7 (36.0)
  Day 11 PM, n=11: number analyzed (Participants) | 11
  Day 11 PM, n=11 | 492.5 (35.2)
  Day 12 AM, n=9: number analyzed (Participants) | 9
  Day 12 AM, n=9 | 451.1 (28.6)
  Day 12 PM, n=11: number analyzed (Participants) | 11
  Day 12 PM, n=11 | 509.5 (33.7)
  Day 13 AM, n=9: number analyzed (Participants) | 9
  Day 13 AM, n=9 | 457.8 (33.9)
  Day 13 PM, n=11: number analyzed (Participants) | 11
  Day 13 PM, n=11 | 506.8 (33.1)
  Day 14 AM, n=11: number analyzed (Participants) | 11
  Day 14 AM, n=11 | 480.5 (30.3)
  Day 14 PM, n=11: number analyzed (Participants) | 11
  Day 14 PM, n=11 | 496.4 (32.1)

32. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for BUD 400 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 8 PM, Day 9 to 14 AM and PM in period 2
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | BUD 400 mcg
Number analyzed (Participants) | 5
Liters per minute
  Day 8 PM | 560.0 (43.3)
  Day 9 AM | 552.0 (40.1)
  Day 9 PM | 560.0 (34.7)
  Day 10 AM | 552.0 (34.9)
  Day 10 PM | 556.0 (30.7)
  Day 11 AM | 562.0 (26.7)
  Day 11 PM | 574.0 (30.4)
  Day 12 AM | 568.0 (29.3)
  Day 12 PM | 578.0 (44.2)
  Day 13 AM | 562.0 (28.1)
  Day 13 PM | 588.0 (37.6)
  Day 14 AM | 586.0 (22.2)
  Day 14 PM | 590.0 (44.6)

33. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for BUD 800 mcg in Period 1
Description: as for outcome 9
Time Frame: Day 15,16, 17, 18, 19, 20, 21 AM and PM in period 1
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | BUD 800 mcg
Number analyzed (Participants) | 11
Liters per minute
  Day 15 AM, n=1: number analyzed (Participants) | 1
  Day 15 AM, n=1 | 610.0 (NA) — NA indicates standard error could not be calculated as only one participant was analyzed.
  Day 15 PM, n=11 | 515.5 (30.1)
  Day 16 AM, n=11 | 494.5 (31.9)
  Day 16 PM, n=11 | 507.3 (34.9)
  Day 17 AM, n=11 | 484.1 (33.4)
  Day 17 PM, n=11 | 505.0 (34.8)
  Day 18 AM, n=11 | 492.7 (33.4)
  Day 18 PM, n=11 | 503.2 (36.4)
  Day 19 AM, n=11 | 483.2 (29.7)
  Day 19 PM, n=11 | 487.7 (38.0)
  Day 20 AM, n=11 | 483.6 (31.7)
  Day 20 PM, n=11 | 517.7 (33.9)
  Day 21 AM, n=11 | 490.5 (27.2)
  Day 21 PM, n=11 | 509.1 (32.9)

34. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for BUD 800 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 15 PM, Day 16, 17, 18, 19, 20, 21 AM and PM in period 2
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | BUD 800 mcg
Number analyzed (Participants) | 5
Liters per minute
  Day 15 PM | 578.0 (32.0)
  Day 16 AM | 568.0 (37.6)
  Day 16 PM | 572.0 (45.3)
  Day 17 AM | 572.0 (27.8)
  Day 17 PM | 558.0 (46.0)
  Day 18 AM | 558.0 (45.8)
  Day 18 PM | 568.0 (53.1)
  Day 19 AM | 572.0 (46.4)
  Day 19 PM | 584.0 (47.3)
  Day 20 AM | 590.0 (37.6)
  Day 20 PM | 590.0 (37.6)
  Day 21 AM | 574.0 (23.5)
  Day 21 PM | 606.0 (38.0)

35. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for BUD 1600 mcg in Period 1
Description: as for outcome 9
Time Frame: Day 22 PM, Day 23,24,25,26,27,28 AM and PM in period 1
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | BUD 1600 mcg
Number analyzed (Participants) | 11
Liters per minute
  Day 22 PM | 506.4 (33.9)
  Day 23 AM | 496.4 (29.8)
  Day 23 PM | 512.7 (32.3)
  Day 24 AM | 498.2 (34.8)
  Day 24 PM | 510.5 (34.9)
  Day 25 AM | 500.5 (32.8)
  Day 25 PM | 514.1 (33.2)
  Day 26 AM | 499.1 (31.3)
  Day 26 PM | 512.3 (35.2)
  Day 27 AM | 491.4 (31.0)
  Day 27 PM | 497.7 (37.3)
  Day 28 AM | 476.8 (27.9)
  Day 28 PM | 526.8 (33.9)

36. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for BUD 1600 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 22 PM, Day 23,24,25,26,27,28 AM and PM in period 2
Population: All subjects Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | BUD 1600 mcg
Number analyzed (Participants) | 5
Liters per minute
  Day 22 PM | 594.0 (47.8)
  Day 23 AM | 578.0 (40.0)
  Day 23 PM | 586.0 (46.4)
  Day 24 AM | 556.0 (37.8)
  Day 24 PM | 556.0 (45.2)
  Day 25 AM | 564.0 (50.6)
  Day 25 PM | 594.0 (45.4)
  Day 26 AM | 584.0 (45.6)
  Day 26 PM | 568.0 (51.1)
  Day 27 AM | 568.0 (52.1)
  Day 27 PM | 584.0 (35.3)
  Day 28 AM | 574.0 (30.1)
  Day 28 PM | 630.0 (46.0)

37. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for BUD 3200 mcg in Period 1
Description: as for outcome 9
Time Frame: Day 29 PM, Day 30, 31,32,33,34,35 AM and PM in period 1
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | BUD 3200 mcg
Number analyzed (Participants) | 10
Liters per minute
  Day 29 PM, n=10 | 493.0 (31.9)
  Day 30 AM, n=10 | 482.0 (33.5)
  Day 30 PM, n=10 | 502.0 (33.3)
  Day 31 AM, n=10 | 482.0 (34.0)
  Day 31 PM, n=10 | 496.0 (32.4)
  Day 32 AM, n=10 | 482.0 (30.1)
  Day 32 PM, n=10 | 488.0 (33.0)
  Day 33 AM, n=10 | 483.0 (29.1)
  Day 33 PM, n=10 | 490.0 (35.0)
  Day 34 AM, n=10 | 489.0 (31.3)
  Day 34 PM, n=9: number analyzed (Participants) | 9
  Day 34 PM, n=9 | 522.2 (33.4)
  Day 35 AM, n=10 | 474.0 (33.8)
  Day 35 PM, n=10 | 488.0 (30.6)

38. Secondary Outcome: Peak Expiratory Flow Rate (PEFR) as a Measure of Safety and Tolerability for BUD 3200 mcg in Period 2
Description: as for outcome 9
Time Frame: Day 29 PM, Day 30, 31,32,33,34,35 AM and PM in period 2
Population: as for outcome 8
Measure: Mean (Standard Error); unit: Liters per minute
Arm/Group | BUD 3200 mcg
Number analyzed (Participants) | 5
Liters per minute
  Day 29 PM, n=5 | 596.0 (43.8)
  Day 30 AM, n=5 | 604.0 (22.7)
  Day 30 PM, n=5 | 586.0 (41.5)
  Day 31 AM, n=4: number analyzed (Participants) | 4
  Day 31 AM, n=4 | 562.5 (33.5)
  Day 31 PM, n=4: number analyzed (Participants) | 4
  Day 31 PM, n=4 | 547.5 (43.8)
  Day 32 AM, n=4: number analyzed (Participants) | 4
  Day 32 AM, n=4 | 592.5 (38.6)
  Day 32 PM, n=4: number analyzed (Participants) | 4
  Day 32 PM, n=4 | 587.5 (18.8)
  Day 33 AM, n=4: number analyzed (Participants) | 4
  Day 33 AM, n=4 | 567.5 (30.3)
  Day 33 PM, n=4: number analyzed (Participants) | 4
  Day 33 PM, n=4 | 565.0 (42.9)
  Day 34 AM, n=4: number analyzed (Participants) | 4
  Day 34 AM, n=4 | 585.0 (38.4)
  Day 34 PM, n=4: number analyzed (Participants) | 4
  Day 34 PM, n=4 | 583.8 (29.6)
  Day 35 AM, n=4: number analyzed (Participants) | 4
  Day 35 AM, n=4 | 577.5 (35.6)
  Day 35 PM, n=4: number analyzed (Participants) | 4
  Day 35 PM, n=4 | 597.5 (38.6)

39. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Vital Signs: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured after participants had rested in supine position for at least 5 minutes. Results are presented treatment wise. No data collected separately for this outcome measure as any abnormal value would be recorded as an Adverse Event.
Time Frame: Up to Week 18
Population: All subjects Population.
Arm/Group | Placebo | FF 25 mcg | FF 100 mcg | FF 200 mcg | FF 400 mcg | FF 800 mcg | FP 50 mcg | FP 200 mcg | FP 500 mcg | FP 1000 mcg | FP 2000 mcg | BUD 100 mcg | BUD 400 mcg | BUD 800 mcg | BUD 1600 mcg | BUD 3200 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

40. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Vital Signs: Pulse Rate
Description: Pulse rate was measured after participants had rested in supine position for at least 5 minutes. Results are presented treatment wise. No data collected separately for this outcome measure as any abnormal value would be recorded as an Adverse Event.
Time Frame: Up to Week 18
Population: All subjects Population
Arm/Group | Placebo | FF 25 mcg | FF 100 mcg | FF 200 mcg | FF 400 mcg | FF 800 mcg | FP 50 mcg | FP 200 mcg | FP 500 mcg | FP 1000 mcg | FP 2000 mcg | BUD 100 mcg | BUD 400 mcg | BUD 800 mcg | BUD 1600 mcg | BUD 3200 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

41. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Vital Signs: Respiratory Rate
Description: Respiratory rate was measured after participants had rested in supine position for at least 5 minutes. Results are presented treatment wise. No data collected separately for this outcome measure as any abnormal value would be recorded as an Adverse Event.
Time Frame: Up to Week 18
Population: All subjects Population.
Arm/Group | Placebo | FF 25 mcg | FF 100 mcg | FF 200 mcg | FF 400 mcg | FF 800 mcg | FP 50 mcg | FP 200 mcg | FP 500 mcg | FP 1000 mcg | FP 2000 mcg | BUD 100 mcg | BUD 400 mcg | BUD 800 mcg | BUD 1600 mcg | BUD 3200 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

42. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Vital Signs: Temperature
Description: Temperature was measured after participants have been rested in supine position for at least 5 minutes. Results are presented treatment wise. No data collected separately for this outcome measure as any abnormal value would be recorded as an Adverse Event.
Time Frame: Up to Week 18
Population: All subjects Population.
Arm/Group | Placebo | FF 25 mcg | FF 100 mcg | FF 200 mcg | FF 400 mcg | FF 800 mcg | FP 50 mcg | FP 200 mcg | FP 500 mcg | FP 1000 mcg | FP 2000 mcg | BUD 100 mcg | BUD 400 mcg | BUD 800 mcg | BUD 1600 mcg | BUD 3200 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

43. Secondary Outcome: Number of Participants With Abnormal Physical Examination
Description: Physical examinations included assessment of the cardiovascular, respiratory, gastrointestinal, skin, abdomen (liver and spleen), and neurological systems. This analysis was planned and data was not collected and captured in the database. Results are presented treatment wise.
Time Frame: Up to Week 18
Population: All subjects Population.
Arm/Group | Placebo | FF 25 mcg | FF 100 mcg | FF 200 mcg | FF 400 mcg | FF 800 mcg | FP 50 mcg | FP 200 mcg | FP 500 mcg | FP 1000 mcg | FP 2000 mcg | BUD 100 mcg | BUD 400 mcg | BUD 800 mcg | BUD 1600 mcg | BUD 3200 mcg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

44. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Hematology Parameters
Description: Blood samples were collected for assessement of following hematology parameters: basophils, eosinophils, Erythrocyte mean corpuscular volume (MCV), hemoglobin, hematocrit, Erythrocyte mean corpuscular hemoglobin (MCH), leukocytes, lymphocytes, monocytes, platelets. Results are presented treatment wise. Only participants with clinically significant abnormal hematology data was reported.
Time Frame: Up to Week 18
Population: All subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | FF 25 mcg | FF 100 mcg | FF 200 mcg | FF 400 mcg | FF 800 mcg | FP 50 mcg | FP 200 mcg | FP 500 mcg | FP 1000 mcg | FP 2000 mcg | BUD 100 mcg | BUD 400 mcg | BUD 800 mcg | BUD 1600 mcg | BUD 3200 mcg
Number analyzed (Participants) | 17 | 20 | 19 | 19 | 18 | 18 | 21 | 20 | 20 | 18 | 17 | 18 | 18 | 18 | 18 | 18
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

45. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Chemistry Parameters
Description: Blood samples were collecte for assessment of following chemistry parametres:Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), albumin, alkaline phosphatase, bilirubin, calcium, creatinine, glucose, direct bilirubin, potassium, protein, sodium, urea. Results are presented treatment wise. Only participants with clinically significant abnormal chemistry data was reported.
Time Frame: Up to Week 18
Population: All subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | FF 25 mcg | FF 100 mcg | FF 200 mcg | FF 400 mcg | FF 800 mcg | FP 50 mcg | FP 200 mcg | FP 500 mcg | FP 1000 mcg | FP 2000 mcg | BUD 100 mcg | BUD 400 mcg | BUD 800 mcg | BUD 1600 mcg | BUD 3200 mcg
Number analyzed (Participants) | 17 | 20 | 19 | 19 | 18 | 18 | 21 | 20 | 20 | 18 | 17 | 18 | 18 | 18 | 18 | 18
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

46. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Urinalysis Parameters
Description: Urine sample were collected to assess following urine parameters: potential of hydrogen (pH), glucose, protein, blood and ketones by dipstick. Results are presented treatment wise. Only participants with clinically significant abnormal urinalysis data was reported.
Time Frame: Up to Week 18
Population: All subjects Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | FF 25 mcg | FF 100 mcg | FF 200 mcg | FF 400 mcg | FF 800 mcg | FP 50 mcg | FP 200 mcg | FP 500 mcg | FP 1000 mcg | FP 2000 mcg | BUD 100 mcg | BUD 400 mcg | BUD 800 mcg | BUD 1600 mcg | BUD 3200 mcg
Number analyzed (Participants) | 17 | 20 | 19 | 19 | 18 | 18 | 21 | 20 | 20 | 18 | 17 | 18 | 18 | 18 | 18 | 18
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

47. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV 1) in Period 1
Description: FEV1 was measured with participants in a sitting position using a calibrated spirometer in accordance with American Thoracic Society (ATS) guidelines using European Respiratory Society (ERS)guidelines for predicted values. Results are presented treatment wise.
Time Frame: Day 1 (pre-dose) in Period 1
Population: All Subjects Population.
Measure: Mean (Standard Error); unit: Liter
Groups:
- Budesonide.: Participants received Participants received BUD Turbuhaler 100 mcg, 400 mcg, 800 mcg, 1600 mcg, 3200 mcg as total daily dose for 7 days.
Arm/Group | Placebo | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide.
Number analyzed (Participants) | 12 | 14 | 15 | 12
Liter | 3.18 (0.151) | 3.02 (0.166) | 3.50 (0.269) | 3.29 (0.274)

48. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV 1) in Period 2
Description: FEV1 was measured with participants in a sitting position using a calibrated spirometer in accordance with ATS guidelines using ERS guidelines for predicted values. Results are presented treatment wise.
Time Frame: Day 1 (pre-dose) in Period 2
Population: All Subjects Population.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD)
Number analyzed (Participants) | 5 | 6 | 6 | 6
Liter | 2.67 (0.482) | 3.44 (0.431) | 2.68 (0.278) | 3.46 (0.257)

49. Secondary Outcome: Forced Vital Capacity (FVC) in Period 1
Description: FVC was measured with participants in a sitting position using a calibrated spirometer in accordance with ATS guidelines using ERS guidelines for predicted values. Results are presented treatment wise.
Time Frame: Day 1 (pre-dose) in Period 1
Population: All Subjects Population.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD)
Number analyzed (Participants) | 12 | 14 | 15 | 12
Liter | 4.55 (0.221) | 4.36 (0.222) | 5.15 (0.287) | 4.70 (0.406)

50. Secondary Outcome: Forced Vital Capacity (FVC) in Period 2
Description: as for outcome 49
Time Frame: Day 1 (pre-dose) in Period 2
Population: All Subjects Population.
Measure: Mean (Standard Error); unit: Liter
Arm/Group | Placebo | Fluticasone Furoate (FF) | Fluticasone Propionate (FP) | Budesonide (BUD)
Number analyzed (Participants) | 5 | 6 | 6 | 6
Liter | 4.11 (0.570) | 4.85 (0.602) | 4.09 (0.386) | 4.90 (0.410)

ADVERSE EVENTS:
Time Frame: Serious adverse events and non-serious adverse events were collected up to 18 weeks.
Description: All subjects Population was used to collect the adverse events.
Arm/Group | Placebo | FF 25 mcg | FF 100 mcg | FF 200 mcg | FF 400 mcg | FF 800 mcg | FP 50 mcg | FP 200 mcg | FP 500 mcg | FP 1000 mcg | FP 2000 mcg | BUD 100 mcg | BUD 400 mcg | BUD 800 mcg | BUD 1600 mcg | BUD 3200 mcg
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/20 | 0/19 | 0/19 | 0/18 | 0/18 | 0/21 | 0/20 | 0/20 | 0/18 | 0/17 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/20 | 0/19 | 0/19 | 0/18 | 0/18 | 0/21 | 0/20 | 0/20 | 0/18 | 0/17 | 0/18 | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 10/17 | 6/20 | 8/19 | 7/19 | 6/18 | 7/18 | 10/21 | 4/20 | 4/20 | 8/18 | 6/17 | 6/18 | 8/18 | 5/18 | 6/18 | 3/18
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | FF 25 mcg (N=20) | FF 100 mcg (N=19) | FF 200 mcg (N=19) | FF 400 mcg (N=18) | FF 800 mcg (N=18) | FP 50 mcg (N=21) | FP 200 mcg (N=20) | FP 500 mcg (N=20) | FP 1000 mcg (N=18) | FP 2000 mcg (N=17) | BUD 100 mcg (N=18) | BUD 400 mcg (N=18) | BUD 800 mcg (N=18) | BUD 1600 mcg (N=18) | BUD 3200 mcg (N=18)
Headache (Nervous system disorders) | 4 (8) | 5 (5) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 2 (3)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 2 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Catheter site bruise (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Catheter site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling jittery (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital discomfort (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keloid scar (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Saliva altered (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinonasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial

DOCUMENTS (2):
  • Study Protocol (2018-04-26): https://cdn.clinicaltrials.gov/large-docs/59/NCT02991859/Prot_000.pdf
  • Statistical Analysis Plan (2019-02-05): https://cdn.clinicaltrials.gov/large-docs/59/NCT02991859/SAP_001.pdf